| INICAL PROTOCOL | Recombinant Botulinum Vaccine<br>A/B (rBV A/B) |
|-------------------|------------------------------------------------|
| CLINICAL PROTOCOL | Protocol<br>rBV A/B-CL-002 |

Protocol rBV A/B-CL-002

# TITLE OF STUDY:

Tolerability and Immunogenicity of a Single 40-µg Dose of Recombinant Botulinum Vaccine A/B (rBV A/B) for the Production of BabyBIG® in Volunteers with Existing Botulinum Immunity.

Date of issue: 05 September 2018

Sponsor:

California Department of Public Health

Infant Botulism Treatment and Prevention Program

850 Marina Bay Parkway, Rm. E-361

Richmond, CA 94804-6403

Phone: 510-231-7600 Fax: 510-231-7609

# Signatures of approval for protocol (Version 1.1)

| Affiliation | Name | Signature | Date |
|---|---|---|---|
| Sponsor-Investigator: | Stephen S. Arnon, M.D.,<br>M.P.H. | Feder C. Annon | 9-5-18 |
| Medical monitor: | John Edward Swartzberg,<br>M.D., F.A.C.P | Sur our ber | 9/5/18 |

CDPH
rBV A/B
Clinical Protocol
IND 015155

# CONFIDENTIAL Recombinant Botulinum Vaccine A/B (rBV A/B) CLINICAL PROTOCOL Protocol rBV A/B-CL-002

Protocol rBV A/B-CL-002

# TITLE OF STUDY:

Tolerability and Immunogenicity of a Single 40- $\mu$ g Dose of Recombinant Botulinum Vaccine A/B (rBV A/B) for the Production of BabyBIG® in Volunteers with Existing Botulinum Immunity.

Date of issue: 05 September 2018

**Sponsor:** California Department of Public Health

**Infant Botulism Treatment and Prevention Program** 

850 Marina Bay Parkway, Rm. E-361

Richmond, CA 94804-6403

Phone: 510-231-7600 Fax: 510-231-7609

# Signatures of approval for protocol (Version 1.1)

| Affiliation Name | | Signature | Date |
|---|---|---|---|
| Sponsor-Investigator: | Stephen S. Arnon, M.D.,<br>M.P.H. | | |
| Medical monitor: | John Edward Swartzberg,<br>M.D., F.A.C.P | | |

rBV A/B
Clinical Protocol IND 015155

This study is to be performed in accordance with Good Clinical Practice, the ethical principles that have their origin in the Declaration of Helsinki, Title 21 of the Code of Federal Regulations, Part 50 (Protection of Human Subjects), Part 56 (Institutional Review Boards), Part 312 (Investigational New Drug Application) and the International Conference on Harmonisation E6 (Guideline for Good Clinical Practice).

Sponsor-Investigator: Stephen S. Arnon, M.D., M.P.H., Chief

Infant Botulism Treatment and Prevention Program

Infectious Diseases Laboratory Branch Division of Communicable Disease Control

Center for Infectious Diseases

California Department of Public Health 850 Marina Bay Parkway, Rm. E-361

Richmond, CA 94804-6403 Phone: 510-231-7600 Fax: 510-231-7609

E-mail: Stephen.Arnon@cdph.ca.gov

Institutional review board: Committee for the Protection of Human Subjects (CPHS)

2020 West El Camino Avenue, Suite 1000

Sacramento, CA 95833 Phone: 916-326-3660 Fax: 916-322-2512

E-mail: cphs-mail@oshpd.ca.gov

Copernicus Group IRB (CGIRB) 5000 Centregreen Way Suite 200

Cary, NC 27513 Phone: 919 465-4310 Fax: 919-465-4311 E-mail: irb@cgirb.com

Medical monitor: John Edward Swartzberg, M.D., F.A.C.P.

Clinical Professor, Emeritus

**UCB-UCSF Joint Medical Program** 

Chair, Editorial Board, UC Berkeley Wellness Letter

University of California, Berkeley

570 University Hall Phone: 510-643-0499 Fax: 510-643-8771 E-mail: jes@berkeley.edu

#### STUDY SYNOPSIS

Name of sponsor company: California Department of Public Health (CDPH)

Name of investigational product: Recombinant Botulinum Vaccine A/B (rBV A/B)

**Names of active ingredients:** Recombinant Botulinum Antigen A and Antigen B adsorbed to 0.2% (wt/vol) Alhydrogel<sup>TM</sup>

Title of study: Tolerability and Immunogenicity of a Single 40-μg Dose of Recombinant Botulinum Vaccine A/B (rBV A/B) for the Production of BabyBIG<sup>®</sup> in Volunteers with Existing Botulinum Immunity

Sponsor Investigator: Dr. Stephen S. Arnon

Number of sites: 2

Study period: 18 months Phase of development: Phase 2

# **Objectives:**

**Immunogenicity:** The immunogenicity objective of this study is to evaluate the effects of a single 40-µg dose of the recombinant botulinum vaccine A/B (rBV A/B) on botulinum toxin type A and type B neutralizing antibody concentration (NAC) over a 12-week period following vaccination in participants who have previously been immunized with pentavalent botulinum toxoid (or pentavalent botulinum toxoid and rBV A/B) for occupational protection.

**Safety:** The safety objective of this study is to obtain safety information during the 12-week study period and at 6 months post-vaccination on the use of rBV A/B in a population of participants previously immunized with pentavalent botulinum toxoid (or pentavalent botulinum toxoid and rBV A/B) for occupational protection.

#### **Exploratory:**

The exploratory objective of this study is to collect source plasma from participants that contains neutralizing antibodies against botulinum toxin type A and type B for the production of BabyBIG.

**Methodology:** This Phase 2, open-label, uncontrolled study designed to evaluate safety, tolerability, and immunogenicity of a single dose of rBV A/B in healthy participants previously immunized with pentavalent botulinum toxoid (or pentavalent botulinum toxoid and rBV A/B) for occupational protection will be conducted to collect source plasma for potential use in the production of BabyBIG and to evaluate safety and immunogenicity of the vaccine in these participants over a 12-week period, with a follow-up safety assessment at 6 months.

The study period is defined as the 12-week period that includes the clinic visits and plasmapheresis visits. The study period will end at Week 4 for participants who opt not to participate in plasmapheresis or who have been determined to be ineligible for plasma donation for the entire study.

**Number of participants (planned):** Up to 50 participants are anticipated to be enrolled.

Name of sponsor company: California Department of Public Health (CDPH)

Name of investigational product: Recombinant Botulinum Vaccine A/B (rBV A/B)

**Names of active ingredients:** Recombinant Botulinum Antigen A and Antigen B adsorbed to 0.2% (wt/vol) Alhydrogel<sup>TM</sup>

#### **Inclusion criteria:**

- Have received pentavalent botulinum toxoid (or pentavalent botulinum toxoid and rBV A/B) for occupational protection under BB-IND-0161 (or BB-IND-0161 and IND 015155)
- Be 18 to 69 years old at the time of consent
- Be healthy and have an acceptable medical history (defined as individuals who are free from significant cardiac, pulmonary, gastrointestinal, hepatic, renal, hematological, neurological, infective, muscular, infectious, rheumatic, immunological, or psychiatric diseases, as determined by medical history over the past 5 years, physical examination, and laboratory tests) that will not interfere with the objectives of the study
- Meet the participant suitability requirements and recommendations for source plasma donors
- If female and of childbearing potential, have a negative pregnancy test at screening and within 24 hours prior to vaccination and must not plan to become pregnant for until after the last plasma donation or until the Week 12 visit (whichever occurs last). Every female participant is considered of childbearing potential unless she has had sterilization surgery or is postmenopausal and has not had a menstrual period for at least 12 months. If the participant is capable of childbearing, she must use a reliable form of contraception approved by the investigator for 30 days before Day 0 through the end of the study. Acceptable forms of contraception include intrauterine device, birth control pills, injectable birth control, implantable birth control device, or removable birth control device or any other United States Food and Drug Administration (U.S. FDA) -approved contraceptive method, or a monogamous relationship with vasectomized partner who has been vasectomized for 6 months or more prior to the participant's study entry, or sexual abstinence.)
- Have the ability to understand the requirements of the study, have provided written informed
  consent as evidenced by signature on an informed consent form approved by the Committee for
  the Protection of Human Subjects, and have agreed to abide by the study restrictions and return for
  the required assessments
- Agree to complete the participant home diary on a daily basis for 7 days post-vaccination, as well as report any adverse events and concomitant medications during the study period
- Have provided written authorization for use and disclosure of protected health information
- Agree not to donate blood or blood products (outside of study procedures) until after the last plasma donation or until the Week 12 visit (whichever occurs last)
- Have personal health insurance

#### **Exclusion criteria:**

- Be pregnant or nursing
- Have a history of laboratory evidence of syphilis, acquired immunodeficiency syndrome, Creutzfeldt-Jakob disease, or infection with human immunodeficiency viruses 1 or 2, human T-cell lymphotropic virus 1, hepatitis B virus, or hepatitis C virus
- Have had a prior severe (Grade 3 or higher) local or severe (Grade 3 or higher) systemic reaction to last immunization with pentavalent botulinum toxoid or a prior severe immediate hypersensitivity reaction or severe systemic reaction to last vaccination on Day 0 with rBV A/B
- Have a known allergy to aluminum compounds, yeast, or other components of the vaccine
- Have donated one or more units of blood or undergone plasmapheresis within 49 days prior to the Vaccination Visit (Day 0)

Name of sponsor company: California Department of Public Health (CDPH)

Name of investigational product: Recombinant Botulinum Vaccine A/B (rBV A/B)

**Names of active ingredients:** Recombinant Botulinum Antigen A and Antigen B adsorbed to 0.2% (wt/vol) Alhydrogel<sup>TM</sup>

- Have received a blood product or immunoglobulin within 6 months of study entry or plans to receive such products during the study period (exclusive of returned red blood cells as part of the plasmapheresis procedure). For participants who choose to donate plasma, this will apply until their last plasma donation or at the Week 12 visit (whichever occurs last)
- Have received licensed nonliving vaccine within 14 days prior to study entry, or licensed live vaccine within 60 days prior to study entry
- Have received investigational products (drugs, biologics, vaccines, or implantable devices) within 60 days prior to study entry or plans to receive experimental products at any time during the study period. For participants who choose to donate plasma, this will apply until their last plasma donation or at the Week 12 visit (whichever occurs last)
- Have received prescription immunosuppressive or immunomodulatory agents, including
  parenteral, inhaled, or oral corticosteroids within 3 months of study entry or plans on receiving
  such therapy at any time during the study period. For participants who choose to donate plasma,
  this will apply until their last plasma donation or at the Week 12 visit (whichever occurs last) with
  the exceptions mentioned below:
  - Participants who have used prescription topical steroids may be enrolled 2 weeks after the therapy is completed
  - o Intra-articular, bursal, or tendon injectable steroids are permitted
  - Any over-the-counter topical steroid use is permitted
  - Ophthalmic and intranasal steroids are permitted
- Have received cytotoxic therapy at any time in the previous 5 years before study entry
- Have an active systemic or recurrent disease that would place the participant at unacceptable risk of injury, require hospitalization, or require surgical intervention (This includes active mental illness or history of mental illness not responsive to treatment.)
- Have a history of alcohol or drug abuse or dependence within 12 months of study entry
- Have past, present, or suspected illicit injection drug use
- Have inflammatory, vasculitic, or rheumatic disease, including systemic lupus erythematosus, polymyalgia rheumatica, rheumatoid arthritis, or scleroderma (Stable osteoarthritis treated with physical therapy and nonsteroidal anti-inflammatory drugs is not an exclusion criterion.)
- Have any acute or chronic neuromuscular or neurologic disorder
- Have clinically confirmed hepatic or renal insufficiency
- Have uncontrolled hypertension, as defined as systolic blood pressure greater than 160 mmHg and diastolic blood pressure greater than 90 mm Hg
- Have moderate to severe asthma, chronic obstructive pulmonary disease, or other significant pulmonary disease
- Have a seizure disorder
- Have moderate or severe illness or oral temperature of 100.4°F or greater within 3 days prior to Vaccination Visit (Day 0)
- Be unsuitable for participation in this study for any reason, as assessed by the investigator

CDPH rBV A/B

IND 015155

Name of sponsor company: California Department of Public Health (CDPH)

Name of investigational product: Recombinant Botulinum Vaccine A/B (rBV A/B)

**Names of active ingredients:** Recombinant Botulinum Antigen A and Antigen B adsorbed to 0.2% (wt/vol) Alhydrogel<sup>TM</sup>

# Test product, dose, and mode of administration:

rBV A/B injections will consist of 40-μg of total antigen (20 μg of Antigen A and 20 μg of Antigen B) adsorbed to 0.2% (wt/vol) Alhydrogel<sup>TM</sup>, in a total dose volume of 0.5 mL. The vaccine will be administered by intramuscular injection in the deltoid muscle, preferably in the nondominant arm.

# Reference therapy, dose, and mode of administration:

No reference therapy will be employed.

**Duration of treatment:** Vaccine administration for all enrolled participants will occur at Day 0, and participants may elect to undergo plasmapheresis up to two times a week for up to 12 weeks, with the final on-site visit at Week 12 ( $\pm$  4 days) and follow-up phone call for safety assessment at Week 26 after vaccination. Participants can elect to continue plasmapheresis up to 14 weeks post-vaccination as long as they continue to meet source plasma donor eligibility requirements.

# Criteria for Evaluation

#### **Populations:**

The immunogenicity population will include all participants who have received the study vaccine at the assigned dosage and for whom at least one post-baseline NAC was collected within 4 weeks of vaccination. For each post-vaccination assessment time point, the per protocol population will include all participants who received the vaccine dose, have a baseline NAC, and have all immunogenicity assessments completed within the protocol-specified timelines (including visit windows) for the time periods summarized and do not have major protocol violations expected to affect immunogenicity. A determination of major protocol violations expected to affect immunogenicity will be done by the sponsor-investigator before reviewing the immunogenicity data for the applicable participant.

# Immunogenicity:

The primary endpoint is as follows:

• The proportion of participants achieving a four times or greater increase in NAC by Week 4 compared with Week 0. A positive response will be defined as achieving this level of increase in at least 50% of the participants for botulinum toxin A and toxin B.

The secondary endpoints are as follows:

- The proportion of participants achieving a two times increase in the area under the plasma concentration-time curve between Week 0 and Week 12 in NAC in comparison to a straight-line extension of the Week 0 NAC to Week 12. A positive response will be defined as achieving this level of increase in at least 50% of the participants for botulinum toxin A and toxin B.
- The proportion of participants achieving a three times or greater increase in NAC by Week 4 compared with Week 0. A positive response will be defined in at least 50% of the participants for botulinum toxin A and toxin B.

# Safety:

Safety analyses will be performed on the safety population, defined as all participants who receive the investigational vaccine. The following analyses will be performed:

Name of sponsor company: California Department of Public Health (CDPH)

Name of investigational product: Recombinant Botulinum Vaccine A/B (rBV A/B)

Names of active ingredients: Recombinant Botulinum Antigen A and Antigen B adsorbed to 0.2% (wt/vol) Alhydrogel<sup>TM</sup>

- Frequency of injection site reactions and systemic reactions in the study population that are characterized as severe or result in a serious adverse event (SAE) during the 0-7 day diary collection period.
- Frequency of injection site reactions and systemic reactions that are characterized as serious adverse events (SAEs).
- Participant incidence of treatment-related SAEs.
- Participant incidence of serious new onset chronic illnesses (NOCIs).
- Clinically significant changes from baseline health that result in an SAE.
- Clinically significant changes in hematology between screening and Week 4 that result in a severe or serious AE.

# Exploratory:

The exploratory endpoint will be the volume of source plasma containing neutralizing antibodies against botulinum toxin type A and type B collected by plasmapheresis for use in BabyBIG manufacture.

Name of sponsor company: California Department of Public Health (CDPH)

Name of investigational product: Recombinant Botulinum Vaccine A/B (rBV A/B)

**Names of active ingredients:** Recombinant Botulinum Antigen A and Antigen B adsorbed to 0.2% (wt/vol) Alhydrogel<sup>TM</sup>

**Study design:** This will be an open-label, uncontrolled study to evaluate the safety and immunogenicity of a single 40-µg intramuscular injection of rBV A/B in participants who were previously immunized with pentavalent botulinum toxoid (or pentavalent botulinum toxoid and rBV A/B) for occupational protection. Participants will receive the rBV A/B injection, and undergo plasmapheresis up to two times per week for up to 14 weeks. Participants will be evaluated for safety and immunogenicity at each study visit with follow-up safety data collected at 6 months. If participants opt not to participate in plasma collections or have been determined to be ineligible to donate plasma for the entire study, they will have a final on-site visit at Week 4 to provide a serum sample for NAC determination and an additional hematology specimen. Participants undergoing plasmapheresis will also have an additional hematology specimen collected at Week 4. Study participants participating in plasma donations will have a final on-site study visit at Week 12. All participants will have a final phone call for safety follow-up at Week 26.

**Experimental procedures:** Participants who meet inclusion criteria and do not meet any exclusion criteria will receive a single rBV A/B injection at Week 0 and will complete a 7-day diary for the Week 1 telephone call. Clinical safety laboratory assessments (serum chemistry, hematology, and urinalysis) will be obtained for all participants at the screening visit. Hematology only will be assessed during the Week 4 visit. Study participants who consent to plasma donation may report to the plasma collection center after the Week 1 visit where they will be assessed by the center for donor eligibility. Once donor eligibility has been confirmed, the participant may choose to donate plasma twice a week for up to 14 weeks.

Safety considerations: Participants will be monitored for serious adverse events after vaccination throughout the 12-week study period and at the Week 26 phone call follow-up. Administration site reactions and systemic reactions will be monitored with a diary provided to collect information, including diameter of any swelling and redness around the injection site and any generalized symptoms between Week 0 and Week 1 in order to determine if any severe reactions or serious adverse events occurred during this 1-week period post-vaccination. All severe local and systemic reactions will be recorded in the electronic case report form (eCRF). Hematology, serum chemistry, and urinalysis specimens will be collected at screening, and repeat hematology at Week 4 for monitoring of any clinically significant changes that result in a severe or serious AE. Clinically significant changes in hematology that result in a severe or serious AE will be recorded on the eCRF. Female participants of childbearing potential will have a urine pregnancy test at screening and again at Week 0 prior to receipt of the vaccine. Source plasma collection will occur for eligible donors at licensed collection locations. If the participant fails to meet donor criteria at any time during the plasmapheresis period, the participant will continue to be followed for serious adverse events according to the study schedule. Participants will be contacted by phone at Weeks 1, 4, and 10. At Week 26, participants will be queried for occurrence of serious adverse events and serious new onset chronic illnesses (NOCIs), which will be recorded by the investigator (or designee) on serious adverse events recording sheets and entered in the eCRF. Vital signs will be monitored at screening, Week 0 (vaccine visit), and at each plasma collection visit.

Name of sponsor company: California Department of Public Health (CDPH)

Name of investigational product: Recombinant Botulinum Vaccine A/B (rBV A/B)

**Names of active ingredients:** Recombinant Botulinum Antigen A and Antigen B adsorbed to 0.2% (wt/vol) Alhydrogel<sup>TM</sup>

**Statistical methods:** The data will be summarized in tables listing the mean, standard deviation or standard error, median, minimum, maximum, and number of participants for continuous data, or in tables listing count and percentage for categorical data, where appropriate.

The immunogenicity parameters are NACs for botulinum toxin type A and type B. These NAC parameters will be analyzed utilizing a validated mouse neutralization assay.

Summaries of local and systemic severe AEs and SAEs related to vaccination (collected in the 7-day diaries) will be produced in tables, by category and severity.

Summaries of clinically significant changes in hematology between screening and Week 4 resulting in a severe or serious AE will be listed.

SAE data will be listed individually and summarized by system organ class and preferred terms and by severity and relatedness.

SAE data of NOCIs will be listed individually and summarized by system organ class and preferred terms and by severity and relatedness.

No formal sample size calculations will be done.

# **TABLE OF CONTENTS**

| | | | Page |
|---|---|---|---|
| TITL | LE OF STUDY: | | 1 |
| 1.0 | INTRODUCTION | | 16 |
| 1.1 | BACKGROUND | | 16 |
| 1.2 | STUDY RATIONALE | | 17 |
| 1.3 | DOSE RATIONALE | | 17 |
| 2.0 | OBJECTIVES | | 19 |
| 2.1 | IMMUNOGENICITY | | 19 |
| 2.2 | SAFETY | | 19 |
| 2.3 | | | |
| 3.0 | | | |
| 3.1 | | | |
| 3.2 | | | |
| J. <b>2</b> | 3.2.1 Inclusion Criteria | | 20 |
| | 3.2.2 Exclusion Criteria | | 22 |
| 3.3 | | | |
| | e ; | | |
| | 3 | | |
| 3.4 | RANDOMIZATION AND BLINDING | | 26 |
| 3.5 | REPLACEMENT OF DROPOUTS | | 26 |
| 4.0 | DRUGS AND DOSAGES | | 27 |
| 4.1 | | N OF INVESTIGATIONAL PRODUCT | |
| 4.2 | DOSING INSTRUCTIONS AND SCHE | DULE | 28 |
| 4.3 | STORAGE AND HANDLING OF INVE | STIGATIONAL PRODUCT | 29 |
| 4.4 | DOSE STOPPING RULES | | 29 |
| | | Rules | |
| 4.5 | • • • • | | |
| 5.0 | | | |
| 5.1 | | ND EVENTS | |
| 5.2 | | NSvs –7 and –1) | |
| | | lasma donors; 4 weeks non-plasma donors) | |
| | | 22, Week 26) | |
| 6.0 | PROCEDURES FOR HANDLING SE | RIOUS ADVERSE EVENTS | 41 |
| 6.1 | DEFINITION OF A SERIOUS ADVERS | SE EVENT | 41 |
| 6.2 | RECORDING SERIOUS ADVERSE EV | ENTS | 42 |

# TABLE OF CONTENTS (continued)

| 6.3 | ASSESS | SMENT OF SEVERITY | 43 |
|---|---|---|---|
| 6.4 | ASSESS | SMENT OF CAUSALITY | 44 |
| 6.5 | EXPEC | TEDNESS OF ADVERSE EVENTS | 46 |
| 6.6 | REPOR | TING OF SERIOUS ADVERSE EVENTS | 46 |
| 6.7 | FOLLO | FOLLOW-UP OF SERIOUS ADVERSE EVENTS | |
| 6.8 | LOCAL | IZED AND SYSTEMIC INJECTION SITE REACTIONS | 48 |
| 6.9 | DATA . | AND SAFETY MONITORING BOARD | 49 |
| 6.10 | PREGN | ANCY | 49 |
| 7.0 | STUDY | OR SITE TERMINATION AND PARTICIPANTDISCONTINUATION | 51 |
| 7.1 | PARTIO | CIPANT DISCONTINUATION | 51 |
| | 7.1.1 | Adverse Event | |
| | 7.1.2 | Intercurrent Illness | |
| | 7.1.3 | Noncompliance | 51 |
| | 7.1.4<br>7.1.5 | Refusal of Investigational Product Administration | |
| 7.2 | | ATURE STUDY OR SITE TERMINATION | |
| <b>8.0</b><br>8.1 | | COLLECTION AND PROCESSING AND STATISTICAL ANALYSIS COLLECTION AND PROCESSING | |
| 8.2 | | STICAL ANALYSIS | |
| | 8.2.1<br>8.2.2 | General Overview | |
| | 8.2.3 | Populations of Interest Baseline Comparability | |
| | 8.2.4 | Immunogenicity Analysis | |
| | 8.2.5 | Safety Analysis | |
| | 8.2.6 | Sample Size | |
| 9.0 | CLINIC | CAL STUDY ADMINISTRATION | 58 |
| 9.1 | | MED CONSENT WITH AUTHORIZATION FOR USE AND DISCLOSURE OF CTED HEALTH INFORMATION | 58 |
| 9.2 | | DOCUMENTATION | |
| 9.2 | 9.2.1 | Investigator Information | |
| | 9.2.1 | Investigators Study Files | |
| | 9.2.3 | Case Report Forms and Source Documentation | |
| | 9.2.4 | Retention of Study Documents | |
| 9.3 | CONFI | DENTIALITY | 60 |
| | 9.3.1 | Data | 60 |
| | 9.3.2 | Participant Anonymity | 60 |
| 9.4 | PROTOCOL COMPLIANCE AND AMENDMENT PROCEDURES | | |
| 9.5 | STUDY | STUDY/DATA MONITOR FUNCTIONS AND RESPONSIBILITY | |
| 10 0 | REFER | FNCES | 62 |

# LIST OF TABLES

| | | Page |
|---|---|---|
| Table 1. | Schedule of Time and Events | 32 |
| Table 2. | Classification of AEs by Severity | 43 |
| Table 3. | Assessment of Causality of Adverse Events | |
| Table 4. | Timeline for Reporting Serious Adverse Events | 47 |
| Table 5. | Protocol Definitions for Severity of Localized Injection Site Reactions | 49 |

# LIST OF FIGURES

| | | Page |
|-----------|--------------------|------|
| Figure 1. | Sample vial label. | 28 |

CDPH rBV A/B IND 015155 CONFIDENTIAL

# Clinical Protocol

# LIST OF APPENDICES

| Appendix A | Code of Federal Regulations Part 640: Additional Standards for Human Blood and Blood |
|---|---|
| | Products |
| Appendix B | Toxicity Tables from Guidance for Industry: Toxicity Grading Scale for Healthy Adult and |
| | Adolescent Participants Enrolled in Preventive Vaccine Clinical Trials |
| Appendix C | Participant Diary |
| Appendix D | Donor History Questionnaire |
| Appendix E | Adverse Event Recording Sheet for Possible Serious Adverse Events (SAEs) |


CDPH rBV A/B Clinical Protocol IND 015155

# LIST OF ABBREVIATIONS

ΑE adverse event

BabyBIG CDPH proprietary name for Botulism Immune Globulin Intravenous (Human) (BIG-IV)

BoNT botulinum neurotoxin

Centers for Disease Control and Prevention CDC **CDPH** California Department of Public Health data and safety monitoring board **DSMB** electronic case report form eCRF

**EDC** electronic data capture ER emergency room **HBV** hepatitis B virus **HCV** hepatitis C virus

human immunodeficiency virus HIV

**ICF** informed consent form

International Conference on Harmonisation **ICH** 

IRB institutional review board investigator site file ISF

MedDRA Medical Dictionary for Regulatory Activities

neutralizing antibody concentration NAC

new onset chronic illness **NOCI** pentavalent botulinum toxoid **PBT** recombinant botulinum vaccine A/B rBV A/B

SAE serious adverse event

treatment-emergent adverse events **TEAE** 

U.S. FDA United States Food and Drug Administration

# 1.0 INTRODUCTION

# 1.1 BACKGROUND

Botulism Immune Globulin Intravenous (Human) (BIG-IV; BabyBIG®) has been demonstrated to significantly shorten hospital stay and improve outcomes in infant botulism patients. BabyBIG is currently produced from antibodies collected from persons with existing botulinum immunity including individuals previously immunized with investigational pentavalent botulinum toxoid (PBT) for occupational protection and/or also boosted with investigational recombinant botulinum vaccine A/B (rBV A/B).

PBT was distributed through the Centers for Disease Control and Prevention (CDC) under BB-IND-0161 for occupational safety. The toxoid was administered to naïve recipients and was also administered as a booster in persons who had been previously immunized. PBT-immunized individuals who have circulating antibodies against botulinum toxin type A and type B are eligible to donate plasma for manufacture of BabyBIG. Donated plasma is fractionated and treated to yield a purified immunoglobulin G product that provides passive immunity to patients with infant botulism.

However, the CDC no longer provides investigational PBT for immunization of laboratory workers at risk for occupational exposure to botulinum serotypes A, B, C, D, and E. Specifically, on the basis of evidence of declining immunogenicity, increasing reactogenicity, and the age of the product, the CDC ceased distribution of PBT after 30 November 2011.<sup>[1]</sup> Thus, a new immunogen against botulinum toxins is needed. A recombinant botulinum vaccine for the toxin serotypes A and B (rBV A/B) has been developed and is being proposed as a replacement vaccine for boosting participants who previously received PBT for occupational protection. This study is the second phase 2 study under IND 15155 being conducted by the California Department of Public Health (CDPH) to determine if rBV A/B will stimulate production of neutralizing antibodies against botulinum toxin types A and B in participants previously immunized with PBT (or PBT and rBV A/B). Participants with a range in neutralizing antibody titers against the toxin types would be candidates for plasma collection for BabyBIG production under IND 15155.

# 1.2 STUDY RATIONALE

This protocol has as its ultimate goal the production of additional lots of the approved orphan drug Botulism Immune Globulin Intravenous (Human), (BIG-IV; BabyBIG<sup>®</sup>) for the treatment of infant botulism. To enable production of BabyBIG, a group of high-titer immunized persons are needed who are willing to donate their hyperimmune plasma as a starting agent (i.e., Source Plasma) for BabyBIG. This protocol is designed to determine botulinum toxin type A and type B neutralizing antibody levels in healthy participants who were previously immunized with PBT (or PBT and rBV A/B) for occupational protection and who receive rBV A/B (or rBV A/B boost). A Phase 2b study conducted by CDPH (rBV A/B-CL-001) demonstrated a single 40-µg dose of rBV A/B was well tolerated and resulted in a significant increase in neutralizing antibodies against botulinum toxins type A and B in participants previously immunized with PBT. The proposed study will continue to evaluate the immunogenicity and safety of a single dose of the rBV A/B vaccine in this previously immunized population. This study design is similar to rBV A/B-CL-001. However, in this study a single 40-µg dose of rBV A/B will be used to stimulate the production of neutralizing antibodies against botulinum toxin type A and type B in participants that are rBV A/B naïve or in participants that volunteered for the rBV A/B-CL-001 clinical trial and received one dose of rBV A/B.

# 1.3 DOSE RATIONALE

An rBV A/B dose of 40-μg of total antigen (20-μg of Antigen A and 20-μg of Antigen B) with Alhydrogel<sup>TM</sup> has been shown in Phase 1 and Phase 2 studies in healthy participants to be effective in stimulating a strong antibody response and has an acceptable safety profile. Most treatment-emergent adverse events (TEAEs) were mild and transient. Furthermore, the safety and immunogenicity of the rBV A/B vaccine in a naïve population was investigated in 372 participants using the same dose level and a three-dose schedule (under BB-IND 11756). A Phase 2b study conducted by CDPH (rBV A/B-CL-001) demonstrated a single 40-μg dose of rBV A/B was well tolerated, and no safety concerns were identified during the study. In addition, the single 40-μg dose resulted in a significant increase in neutralizing antibodies against botulinum toxin types A and B in participants previously immunized with PBT. Therefore, the proposed dose in this study is expected to have an acceptable safety profile and be effective in stimulating

CDPH rBV A/B IND 015155 CONFIDENTIAL

Clinical Protocol

antibody response in persons previously immunized with PBT for occupational protection.

# 2.0 OBJECTIVES

# 2.1 IMMUNOGENICITY

The immunogenicity objective of this study is to evaluate the effects of a single 40-µg dose of rBV A/B on the botulinum toxin type A and type B neutralizing antibody concentration (NAC) over a 12-week period following vaccination in participants previously immunized with PBT (or PBT and rBV A/B) for occupational protection.

# 2.2 SAFETY

The safety objective of this study is to obtain safety information during the 12-week study period and at 6 months post-vaccination on the use of rBV A/B in a population of participants previously immunized with PBT (or PBT and rBV A/B) for occupational protection.

# 2.3 EXPLORATORY

The exploratory objective of this study is to collect source plasma from participants that contains neutralizing antibodies against botulinum toxin type A and type B for the production of BabyBIG.

# 3.0 STUDY DESIGN

# 3.1 BASIC DESIGN CHARACTERISTICS

This will be an open-label, uncontrolled study to evaluate the safety and immunogenicity of a single intramuscular injection of 40-µg of rBV A/B in participants who were previously immunized with PBT (or PBT and rBV A/B) for occupational protection. Participants will receive the rBV A/B injection, and may elect to undergo plasmapheresis at a maximum of two times per week up to 12 weeks. Participants can continue plasmapheresis up to 14 weeks as long as they continue to meet source plasma donor acceptance criteria. Participants will be evaluated for safety and immunogenicity at each study visit with longer-term follow-up safety data collected at 6 months.

The study period is defined as the 12-week period that includes the clinic visits and plasmapheresis visits. The study period will end at Week 4 for participants who opt not to participate or who have been determined to be ineligible for donation for the entire study. Participants undergoing plasmapheresis will also have an additional hematology specimen collected at Week 4. Study participants participating in plasma donations will have a final on-site study visit at Week 12. All participants will have a final phone call for safety follow-up at Week 26.

# 3.2 STUDY POPULATION

For this study, up to 50 participants are anticipated to be enrolled. Eligibility will be established by the investigator(s) on the basis of the inclusion and exclusion criteria.

# 3.2.1 Inclusion Criteria

To be considered eligible to participate in this study, a participant must meet the inclusion criteria listed below:

- Have received pentavalent botulinum toxoid (or pentavalent botulinum toxoid and rBV A/B) for occupational protection under BB IND 0161 (or BB-IND-0161 and IND 015155)
- 2. Be 18 to 69 years old at the time of consent

- 3. Be healthy and have an acceptable medical history (defined as individuals who are free from significant cardiac, pulmonary, gastrointestinal, hepatic, renal, hematological, neurological, infective, muscular, infectious, rheumatic, immunological, or psychiatric diseases, as determined by medical history over the past 5 years, physical examination, and laboratory tests) that will not interfere with the objectives of the study
- 4. Meet the participant suitability requirements and recommendations for source plasma donors outlined in Appendix A.
- 5. If female, and of childbearing potential, have a negative pregnancy test at screening and within 24 hours prior to vaccination and must not plan to become pregnant until after the last plasma donation or until the Week 12 visit ([whichever occurs last]. Every female participant is considered of childbearing potential unless she has had sterilization surgery or is postmenopausal and has not had a menstrual period for at least 12 months.) If the participant is capable of childbearing, she must use a reliable form of contraception approved by investigator for 30 days before Day 0 through the end of the study. Acceptable forms of contraception include intrauterine device, birth control pills, injectable birth control, implantable birth control device, or removable birth control device or any other United States Food and Drug Administration (U.S. FDA) -approved contraceptive method, or a monogamous relationship with vasectomized partner, who has been vasectomized for 6 months or more prior to the participant's study entry, or sexual abstinence.)
- 6. Have the ability to understand the requirements of the study, have provided written informed consent as evidenced by signature on an informed consent form (ICF) approved by the Committee for the Protection of Human Subjects, and have agreed to abide by the study restrictions and to return for the required assessments
- 7. Agree to complete the participant home diary on a daily basis for 7 days post-vaccination, as well as to report any adverse events and concomitant medications during the study period
- 8. Have provided written authorization for use and disclosure of protected health information

9. Agree not to donate blood or blood products (outside of study procedures) until after the last plasma donation or until the Week 12 visit (whichever occurs last)

10. Have personal health insurance

# 3.2.2 Exclusion Criteria

To be eligible for entry into the study, the participant must not meet any of the exclusion criteria listed below:

- 1. Be pregnant or nursing
- 2. Have a history of laboratory evidence of syphilis, acquired immunodeficiency syndrome, Creutzfeldt-Jakob disease, or infection with human immunodeficiency viruses (HIV) 1 or 2, human T-cell lymphotropic virus 1, hepatitis B virus (HBV), or hepatitis C virus (HCV)
- 3. Have had a prior severe (Grade 3 or higher) local or severe (Grade 3 or higher) systemic reaction to last immunization with pentavalent botulinum toxoid or a prior severe immediate hypersensitivity reaction or severe systemic reaction to last vaccination on Day 0 with rBV A/B
- 4. Have known allergy to aluminum, yeast, or other components of the vaccine
- 5. Have donated one or more units of blood or undergone plasmapheresis within 49 days of the Vaccination Visit (Day 0)
- 6. Have received blood product or immunoglobulin within 6 months prior to study entry or plans to receive such products during the study period (exclusive of returned red blood cells as part of the plasmapheresis procedure). For participants who choose to donate plasma, this will apply until their last plasma donation or at the Week 12 visit (whichever occurs last)
- 7. Have received licensed nonliving vaccine within 14 days prior to study entry, or licensed live vaccine within 60 days prior to study entry

- 8. Have received investigational products (drugs, biologics, vaccines, or implantable devices) 60 days prior to study entry or plans to receive experimental products at any time during the study period. For participants who choose to donate plasma, this will apply until their last plasma donation or at the Week 12 visit (whichever occurs last)
- 9. Have received prescription immunosuppressive or immunomodulatory agents, including parenteral, inhaled, or oral corticosteroids within 3 months of study entry or plans on receiving such therapy at any time during the study period [For participants who choose to donate plasma, this will apply until their last plasma donation or at the Week 12 visit (whichever occurs last)], with the exceptions mentioned below
  - Participants who have used prescription topical steroids may be enrolled
     2 weeks after the therapy is completed
  - Intra-articular, bursal, or tendon injectable steroids are permitted
  - Any over-the-counter topical steroid use is permitted
  - Ophthalmic and intranasal steroids are permitted
- 10. Have received cytotoxic therapy at any time in the previous 5 years before study entry
- 11. Have an active systemic or recurrent disease that would place the participant at unacceptable risk of injury, require hospitalization, or require surgical intervention (This includes active mental illness or history of mental illness not responsive to treatment.)
- 12. Have a history of alcohol or drug abuse or dependence within 12 months of study entry
- 13. Have past, present, or suspected illicit injection drug use
- 14. Have inflammatory, vasculitic, or rheumatic disease, including systemic lupus erythematosus, polymyalgia rheumatica, rheumatoid arthritis, or scleroderma

- 15. Have any acute or chronic neuromuscular or neurologic disorder
- 16. Have clinically confirmed hepatic or renal insufficiency
- 17. Have uncontrolled hypertension, as defined a systolic blood pressure greater than 160 mmHg and diastolic blood pressure greater than 90 mmHg
- 18. Have moderate to severe asthma, chronic obstructive pulmonary disease, or other significant pulmonary disease
- 19. Have a seizure disorder
- 20. Have moderate or severe illness or oral temperature of 100.4°F or greater within 3 days of Vaccination Visit (Day 0)
- 21. Be unsuitable for participation in this study for any reason, as assessed by the investigator

# 3.3 ENDPOINTS

# 3.3.1 Immunogenicity

The primary immunogenicity endpoint is the proportion of participants achieving a four times or greater increase in NAC by Week 4 compared with Week 0. A positive response will be defined as achieving this level of increase in at least 50% of the participants for botulinum toxin type A and type B.

The secondary immunogenicity endpoints are as follows:

 The proportion of participants achieving a two times increase in the area under the plasma concentration-time curve between Week 0 and Week 12 in NAC in comparison to a straight-line extension of the Week 0 NAC to Week 12. A positive response will be defined as achieving this level of increase in at least 50% of the participants for botulinum toxin type A and type B.

• The proportion of participants achieving a three times or greater increase in NAC by Week 4 compared with Week 0. A positive response will be defined as achieving this level of increase in at least 50% of the participants for botulinum toxin type A and type B.

# **3.3.2 Safety**

Primary safety endpoints will be collected over a 12-week period and will be as follows:

- Frequency of injection site reactions and systemic reactions that are characterized as severe during the 0-7 day diary collection period.
- Frequency of injection site reactions and systemic reactions that are characterized as serious adverse events (SAEs) [Definitions for local injection site reactions are in Section 6.9 and systemic reactions are located in Appendix B. Definition of SAE is located in Section 6.1]
- Participant incidence of treatment-related serious adverse events (Adverse event toxicity tables are located in Appendix B)
- Participant incidence of serious NOCIs
- Clinically significant changes from baseline health resulting in serious adverse events
- Clinically significant changes in hematology between screening and Week 4 resulting in severe or serious adverse events

# 3.3.3 Exploratory

The exploratory endpoint will be the volume of source plasma containing neutralizing antibodies against botulinum toxin type A and type B collected by plasmapheresis for use in BabyBIG manufacture.

CONFIDENTIAL CDPH rBV A/B Clinical Protocol IND 015155

# 3.4 RANDOMIZATION AND BLINDING

There will be no randomization or blinding of participants for safety assessments in this study.

# 3.5 REPLACEMENT OF DROPOUTS

Dropouts will not be replaced in this study.

# 4.0 DRUGS AND DOSAGES

# 4.1 IDENTIFICATION AND DESCRIPTION OF INVESTIGATIONAL PRODUCT

# 4.1.1 Investigational Product

rBV A/B is manufactured by DynPort Vaccine Company LLC, a GDIT Company (Frederick, Maryland). The procedure used to manufacture the active ingredient of rBV A/B is described below.

The recombinant botulinum neurotoxin antigens are expressed from synthetic genes encoding the carboxy-terminal region of the botulinum neurotoxins (BoNT) heavy-chains [rBoNT(Hc)] of BoNT/A and BoNT/B, designated Antigen A and Antigen B. These fragments are from the binding domain of the heavy-chain and do not have neurotoxic activity. Antigen A and Antigen B are expressed in the methylotrophic yeast *Pichia pastoris* as 50 kDa and 52 kDa proteins, respectively. Antigen A is derived from the BoNT/A1 expressed by *Clostridium botulinum* strain NCTC 2916 (Group I, proteolytic), and Antigen B is derived from BoNT/B1 expressed by *C. botulinum* strain Danish (Group I, proteolytic). These proteins have been expressed individually by using a methanol induction system from synthetic genes introduced into *P. pastoris*. The bulk antigens were manufactured at high purity (each antigen purified drug substance is >95% pure), formulated and combined in a 1:1 ratio based on mass (in micrograms) to produce the final drug product.

The formulation used for this study will have 40 micrograms (μg) total antigen (20 μg Antigen A and 20 μg Antigen B) with 100 mM sodium chloride, 15 mM sodium phosphate, and 50 mM sodium acetate with Alhydrogel<sup>TM</sup> (0.2% weight per volume) balanced to a pH of 5.5 for a total dose volume of 0.5 mL.


CDPH
rBV A/B
Clinical Protocol

IND 015155

# 4.1.2 Labeling

Each vial in Lot D1200138 will be labeled as shown in Figure 1.

Figure 1. Sample vial label.



# 4.2 DOSING INSTRUCTIONS AND SCHEDULE

Participants will receive a 0.5 mL intramuscular injection of rBV A/B in the deltoid muscle, preferably in the nondominant arm. The injection will be administered by the investigator or delegated site personnel. Site personnel will document the time of the injection in the electronic case report form (eCRF). Each vial should be visually inspected for particulate matter, discoloration, signs of adulteration, or contamination before administration. If the product appears discolored or has visible particulate matter, it should not be used and both the study monitor and principal investigator should be notified. If the investigational product in the vial is suspect, it should not be dispensed or administered. Instead, a new dose should be obtained, inspected, and the dose withdrawn then administered. The occurrence of such an event should be recorded in the ISF (investigator site file).

Each vial will be prepared by swirling gently immediately before use. Approximately 0.5 to 0.6 mL of investigational product will be drawn into a sterile, 1 mL latex-free tuberculin syringe (Becton Dickinson & Co.) or equivalent with a sterile, 21-gauge, 1-inch BD PrecisionGlide<sup>TM</sup> Needle (Becton Dickinson & Co.) or equivalent. To ensure a full dose is able to be drawn from each vial, the vial may need to be inverted with the bevel of the needle inserted just above the rubber stopper. The date, time, and administrator's initials will be recorded in the participant's source record and on the Investigational Product Accountability Log upon administering the investigational product to the participant. In addition, the

site of vaccination (e.g., deltoid muscle of left arm) will be recorded in the participant's source medical record.

# 4.3 STORAGE AND HANDLING OF INVESTIGATIONAL PRODUCT

All vials will be stored at 2°C to 8°C (35.6°F to 46.4°F) in a secure storage location. The refrigerator temperature will be recorded continuously and monitored daily. The investigational product must not be frozen. A copy of the temperature logs for the storage refrigerator must be filed in the site study files to document appropriate storage conditions.

The principal investigator must ensure that accurate records of receipt of all vaccine, including date of receipt, are maintained throughout the study. In addition, accurate records must be kept regarding when and how much vaccine was used.

Study personnel must not destroy or throw away any vial of vaccine, including empty, damaged, or partially used ones. At the completion of the study, to satisfy regulatory requirements regarding drug accountability, all vaccine will be reconciled and the study monitor will verify that the remaining vials have been either returned to designee as determined by the sponsor-investigator or destroyed following the sponsor-investigator's instructions.

# 4.4 DOSE STOPPING RULES

# 4.4.1 Individual Participant Stopping Rules

Because only one dose of vaccine is administered per participant, there will be no individual participant stopping rules to preclude further vaccination.

Participants who develop a Grade 3 (or higher) immediate hypersensitivity reaction to the vaccine will be counselled by the investigator that future exposure to rBV A/B would not be advisable.

# 4.4.2 Study Stopping Rules

For this study, the following are the dose stopping rules; and, if they occur, all dosing will stop, the DSMB (Section 6.10) will convene, review the data collected, and make a recommendation for continued dosing.

- If any participant has an SAE (see Section 6.1 for a definition) considered possibly, probably, or definitely related to the vaccine
- Two or more participants with a Grade 3 (severe) or higher similar hematologic abnormality, considered possibly, probably or definitely related to the vaccine
- Two or more participants with neuromuscular AEs considered possibly, probably or definitely related to the vaccine

If the DSMB determines that an SAE was a vaccine-related SAE, then the sponsor-investigator will provide the DSMB's recommendation along with the SAE report to the FDA and seek the Agency's guidance on resuming the study.

# 4.5 CONCOMITANT MEDICATIONS

There are no restrictions on concomitant medications for the treatment of adverse events. All prior and current medications taken within 60 days prior to Screening will be collected and recorded in the eCRF. Concomitant medications will be queried for at each study visit. Any concomitant medication used to treat a severe injection site or systemic reaction from Week 0-1 as well as any SAEs or serious NOCIs throughout the study (through Week 26) will be recorded in the eCRF.

Enrolled participants should not receive licensed preparations of botulinum toxin A or B used to treat spastic disorders because they are already immune to the therapeutic benefits.

Enrolled participants should not receive any additional vaccines during the study period. For participants who choose to donate plasma, this will apply until their last plasma donation or at the Week 12 visit (whichever occurs last).

Participants should not receive prescription immunosuppressive agents, including corticosteroids (systemic and inhalational), during the study period. For participants who choose to donate plasma, this will apply until their last plasma donation or at the Week 12 visit (whichever occurs last). Intra-articular, bursal or tendon injectable steroids are permitted. Ophthalmic and intranasal steroids are permitted. Over-the counter topical steroids are permitted.

# 5.0 EXPERIMENTAL PROCEDURES

# 5.1 OVERVIEW: SCHEDULE OF TIME AND EVENTS

For this clinical trial there is a 7-day screening period (Days -7 to -1) in which participant eligibility will be determined. Participants will enter either a 4-week (non-plasma donors) or a 12-week (plasma donors) treatment period in which a single rBV A/B injection will be administered on Day 0 to stimulate the production of antibodies against botulinum toxin type A and type B. Participants will be able to donate plasma starting 1 week after injection with rBV A/B at a frequency of up to two times a week, for up to 12 weeks with the possibility of extending the donation times up to 14 weeks post-vaccination in accord with FDA plasma donation regulations and guidelines.<sup>[2]</sup> NAC sample collections are required for all participants at Week 0 and Week 4. NAC sample collection is required for plasma donors with each donated unit. Safety assessments for non-plasma donors are scheduled on Week 0, Week 1 (by phone), and Week 4 (final on-site visit). Safety assessments for plasma donors are at Week 0 with follow-up phone calls at Weeks 1, 4 and 10, and a final on-site study visit at Week 12 to assess general health status and query for the interim occurrence of any SAEs or NOCIs. All participants will have a final phone call for safety follow-up at Week 26. Concomitant medications will be queried for at each study visit. Any concomitant medication used to treat a severe injection site or systemic reaction from Week 0-1 as well as any SAEs or serious NOCIs throughout the study will be recorded in the eCRF.

The schedule of events is presented in Table 1.

Table 1. Schedule of Time and Events

| | | | | Study Period | | | | |
|---|---|---|---|---|---|---|---|---|
| Measurements/Evaluations | Screening | Vaccination<br>Visit | Telephone<br>Call | Telephone Call | Telephone<br>Call | Plasmapheresis | Final Study Visit | Follow-up Call |
| | Day -7 to -1 | Week 0,<br>Day 0 | Week 1 <sup>a</sup> | Week 4 <sup>a, b</sup> | Week 10 <sup>a</sup> | Week 2- 14 <sup>c</sup> | Week 12 <sup>d</sup> | Week 26 <sup>e</sup> |
| Informed consent | X | | | | | X <sup>f</sup> | | |
| Physical examination | X | | | | | X <sup>g</sup> | | |
| Medical history | X | | | | | | | |
| Prior medication history | X | | | | | | | |
| Urine pregnancy test | X | $X^h$ | | | | | X | |
| Inclusion/exclusion criteria | X | X | | | | | | |
| Vital signs | X | $X^{i}$ | | | | X | | |
| Informed consent for plasma | X | | | | | | | |
| collection | | | | | | | | |
| HIV, HBV, and HCV tests <sup>j</sup> | | | | | | X | | |
| Hematology | $X^k$ | | | $X^{l}$ | | | | |
| Serum chemistry | $X^k$ | | | | | | | |
| Urinalysis | $X^k$ | | | | | | | |
| NAC sample collection | | $X^{m}$ | | X <sup>n</sup> | | X | X | |
| Plasmapheresis <sup>o</sup> | | | | | | X | | |
| rBV A/B injection | | X | | | | | | |
| Injection site evaluation | | $X^p$ | | X | | | X | |
| Diary distribution <sup>q</sup> | | X | | | | | | |
| Diary review | | | X | | | | | |
| Serious adverse event | | X | X | X | X | | X | X |
| collection <sup>r</sup> | | | | | | | | |
| Concomitant medication | X <sup>t</sup> | | Xs | Xs | $X^{s}$ | | Xs | Xs |
| information | | | V | 37 | 37 | | | V |
| Phone call | | | X | X | X | | | X |

HBV = hepatitis B virus; HCV = hepatitis C virus; HIV = human immunodeficiency virus; NAC = neutralizing antibody concentration; rBV A/B = recombinant botulinum vaccine A/B. a. Week 1, Week 4, and Week 10 Follow-up Calls must occur with ±3 days of the scheduled time.

b. Final Study Visit will be an on-site visit at Week 4 for participants who opt not to participate or who have been determined to be ineligible for donation for the entire study. All final assessments occurring at Week 12 will occur at Week 4 for these participants.

c. Extension of plasmapheresis for up to 14 weeks is optional

Clinical Protocol

d. Final on-site Study Visit must occur within  $\pm$  7 days of the scheduled time.

- e. Final follow-up call for safety must occur within ±1 week of the scheduled time.
- f. Plasmapheresis-specific informed consent formed will be signed at the source plasma center.
- g. Physical examination will be performed as part of source plasma donor screening at the plasma collection center
- h. Female participants of childbearing potential must have a negative pregnancy test within 24 hours prior to vaccination.
- i. Participants will have vital signs taken twice at Visit 1: prior to injection, and 30 minutes (± 5 minutes) after receiving the injection.
- j. HIV, HBV, and HCV tests will be performed on each donated source plasma unit
- k. Results from screening tests must be available before Vaccination Visit
- 1. Study participants will go to central lab or plasma center for this draw (not an on-site visit).
- m. Baseline NAC sample must be collected before rBV A/B injection and before plasmapheresis
- n. Participants not donating plasma must go to site for NAC collection within ±3 days of the scheduled time.
- o. May occur up to twice a week for up to 14 weeks (if hemoglobin and total protein remain within acceptable range) following vaccination with rBV A/B.
- p. At this visit, participants will be monitored for at least 30 minutes after injection for a possible reaction.
- q. In the diaries, participants record adverse events in order to determine SAE, oral temperature and injection site information.
- r. Only serious adverse events and new onset chronic illnesses are to be queried for and collected
- s.. All concomitant medication used to treat a severe injection site or systemic reaction from Week 0-1 as well as any SAEs or serious NOCIs throughout the study (through Week 26) will be queried for and collected.
- t. All prior and current medications taken within 60 days prior Screening will be queried for and collected.

rBV A/B
Clinical Protocol IND 015155

# 5.2 MEASUREMENTS AND EVALUATIONS

This section details the visits that occur during the study and the assessments that are conducted at each visit. Details of the assessments performed during the study are provided at the visit at which they are first performed.

NAC determinations will be performed at Battelle Biomedical Research Center (Columbus, Ohio) using a fully validated mouse neutralization assay for all NAC determinations in the BabyBIG program.

# 5.2.1 Screening Period (between Days –7 and –1)

Before the initiation of screening assessments, the participant will be given a complete explanation of the purpose and evaluations of the study. Subsequently, the participant must sign and receive a copy of the institutional review board (IRB) approved ICF (Section 9.1) that includes authorization for use and disclosure of protected health information (Section 9.1). Once the ICF has been obtained, the baseline screening assessments will be performed and the eligibility of the participant will be determined. The participant will be assigned a participant number once the ICF is signed. A separate plasmapheresis ICF must be obtained for participants donating plasma.

Screening must occur between 1 and 7 days before Visit 1 (i.e. Vaccination Visit [Day 0]). The following evaluations will be performed to assess the participant's eligibility for the study:

- Medical history
- Physical examination, including weight and height; head, eyes, ears, nose, and throat; respiratory; cardiovascular; gastrointestinal; extremities; skin; neurologic and mental status evaluation
- Vital signs (temperature, blood pressure, heart rate, and respiratory rate)
- Urine pregnancy test (If positive, perform confirmatory blood test.)
- Listing of prior and current medications for past 60 days
- Hematology panel:

CONFIDENTIAL CDPH rBV A/B Clinical Protocol IND 015155

- Hemoglobin

- White blood cell count (with absolute count lymphocytes, neutrophils, eosinophils)
- Platelets

# • Serum chemistry panel:

- Glucose
- Blood urea nitrogen
- Creatinine
- Alanine aminotransferase
- Calcium
- Potassium
- Aspartate aminotransferase
- Alkaline phosphatase
- Bilirubin
- Urinalysis (dipstick testing of clean-catch sample)
  - Protein
  - Glucose
  - Blood
  - Ketones
  - Leukocyte esterase

The investigator may use clinical judgment when determining the clinical relevance of laboratory parameter findings throughout the study. Depending on study criteria, the medical monitor maybe consulted before enrollment about a potential participant with abnormal laboratory values. Guidance on abnormal laboratory values is given in Appendix B.

Total blood volume collected at this visit will be 10 mL (5 mL each for the hematology and serum chemistry). Total urine volume collected will be approximately 30 mL for the urinalysis and urine pregnancy test.

# 5.2.2 Treatment Period (12 weeks, plasma donors; 4 weeks non-plasma donors)

During this period, participants will have visits and phone calls as outlined below. If the participant discontinues, effort should be made to conduct the assessments of the Week 12 visit or end-of-study visit for the participant at Week 4.
# 5.2.2.1 Vaccination Visit (Week 0, Day 0)

During this visit, the following activities will occur:

- Review of baseline health assessment and inclusion and exclusion criteria
- Urine pregnancy test for female participants of childbearing potential, performed within 24 hours preceding receipt of the study vaccine.
- Collection of 20 mL of blood to determine NAC
- Vital signs (temperature, blood pressure, heart rate, and respiratory rate) assessed before the injection and 30 minutes ( $\pm$  5 minutes) after the injection
- Injection of rBV A/B
- Participant monitored for at least 30 minutes after injection for localized and systemic reactions, including vital signs taken at the end of the 30-minute period
- Reaction Recording Sheet Participant Home Diary distributed to the participant to record injection site information and systemic reactions, if any, as well as concomitant medications taken for potential reactions (copy of diary is in Appendix C)
- Adverse Event Recording Sheet for Identification of Possible Serious Adverse
  Events distributed to the participant to record adverse events, for 7 days (copy
  of recording sheet is in Appendix E)

Total blood volume collected at this visit will be 20 mL for NAC.

# 5.2.2.2 Plasma Donation Period (up to 14 weeks)

After receiving the rBV A/B vaccination, the participant may participate as a source plasma donor if they choose. A screening physical exam will be performed at the plasma collection center. Donor eligibility will be determined at the sponsor-approved, licensed source plasma collection center. Once donor eligibility has been confirmed, the participant may begin donating plasma 1 week after vaccination up to twice a week for the next 12 weeks, with the possibility of continuing for up to 14 weeks, consistent with FDA plasma donation regulations and guidelines.<sup>[2]</sup>

During the first visit to the plasma collection center, the following activities will occur:

- Brief physical examination by a licensed physician or otherwise authorized designee at the plasma collection center (the medical exam for plasmapheresis is repeated on an annual basis)
- Measurement of vital signs (temperature, blood pressure, heart rate, and respiratory rate)
- Obtaining informed consent for plasma donation and procedures
- Completion of donor history questionnaire (Appendix D)
- Finger prick for hemoglobin measurement and total serum protein measurement
- Approximately 10 mL of whole blood collected for atypical antibody measurements, serologic test for syphilis, and serum protein electrophoresis at 4-month intervals
- Obtaining 20 mL whole blood by side sample collections for NAC determination
- Plasma donation (takes approximately 1 to 1.5 hours) per the donation site's procedures
- Each donated unit will be tested for infectious markers using nucleic acid testing

During each subsequent visit to the plasma collection center, the following activities will occur:

- Completion of the donor history questionnaire
- Measurement of vital signs (temperature, blood pressure, heart rate, and respiratory rate)
- Finger prick for hemoglobin measurement and total serum protein measurement
- Obtaining 20 mL whole blood by side sample collections for NAC determination

CDPH rBV A/B

IND 015155

Plasma donation (takes approximately 1 to 1.5 hours) per the donation site's

Clinical Protocol

Each donated unit will be tested for infectious markers using nucleic acid testing

Samples for NAC determination will be obtained before plasma collection. The source plasma from plasmapheresis will be retained and is eligible for use in the production of BabyBIG.

Participants will be able to complete plasma donations at a maximum of twice a week up to 12 weeks after the rBV A/B injection, with the possibility of further donation time up to 14 weeks consistent with FDA plasma donation regulations and guidelines for hemoglobin and total protein. At 4-month intervals, the participant will have an additional tube of whole blood drawn at the plasmapheresis center for atypical antibody measurements and serum protein electrophoresis. These additional blood draw results will not be included among the study data.

#### 5.2.2.3 **Telephone Call (Week 1)**

procedures

Study personnel will call participants at Week 1 ( $\pm$  3 days) to review the Reaction Recording Sheet – Participant Home Diary injection site and systemic reactions, as well as any potential SAEs occurring over the past week and any NOCIs and concomitant medications. Study personnel should inquire about participants overall well-being and any concomitant medications. Participants should use the provided Adverse Event Recording Sheet for Identification of Possible Serious Adverse Events form (Appendix E) between phone calls to assist during the inquiry. The information recorded by the delegated site personnel during the phone call will serve as the source documentation.

#### 5.2.2.4 Week 4 Visit and Laboratory Draws

Participants not participating in plasma donation must return to the site at Week 4  $(\pm 3 \text{ days})$  for their final study visit. During this visit, the following activities will occur:

Injection site inspection

- Review of serious adverse events
- Review of any new onset chronic illnesses
- Collection of concomitant medication information, if any
- Collection of 20 mL of blood to determine NAC
- Urine pregnancy test for female participants of childbearing potential
- Repeat of hematology conducted at screening (Section 5.2.1)
- Completion of final on-site study record

Total blood volume collected at this visit will be 25 mL (20 mL for NAC and 5 mL for hematology). Total urine volume collected will be approximately 10 mL for the urine pregnancy test.

All participants continuing in the study will go to a central lab or plasma center (not on site) for hematology.

# 5.2.2.5 Telephone Calls (Weeks 4 and 10)

Study personnel will call plasma donating participants at Weeks 4 ( $\pm$  3 days) and 10 ( $\pm$  3 days) to inquire about participants overall well-being, SAEs, if any, that occurred since the last visit or phone call, any concomitant medication used, any NOCIs, any AEs that increased in severity and injection site or systemic reactions. SAEs, including serious NOCIs, serious injection site or systemic reactions and concomitant medication used as treatment will be recorded in the eCRF.

### 5.2.2.6 Week 12 Visit

For all participants participating in plasma donation, the final on-site study visit must occur within 1 week of Week 12. During this visit, the following activities will occur:

- Injection site inspection
- Review of serious adverse events or serious NOCIs

CDPH rBV A/B IND 015155

- Collection of concomitant medication information used for treatment of any SAEs or serious NOCIs, if any
- Collection of 20 mL of blood to determine NAC
- Urine pregnancy test for female participants of childbearing potential
- Completion of final on-site study record

Total blood volume collected at this visit will be 20 mL for NAC determinations. Total urine volume collected will be approximately 10 mL for the urine pregnancy test.

# 5.2.3 Final Study Follow-up (Day 182, Week 26)

Within 1 week of Week 26, site personnel will contact the participant by phone to assess the participant's general health status. Interim occurrence of any SAEs or serious NOCIs will be queried for and recorded. Any concomitant medications used to treat SAEs or serious NOCIs will be recorded and entered in the eCRF.

### 6.0 PROCEDURES FOR HANDLING SERIOUS ADVERSE EVENTS

### 6.1 DEFINITION OF A SERIOUS ADVERSE EVENT

In this clinical trial, a *serious adverse event* is defined as an AE that meets any of the following criteria:

- Results in death
- Is life-threatening

The term *life-threatening* in the definition of an SAE refers to an event in which the participant was at risk of death at the time of the event. *Life-threatening* does not refer to an event that hypothetically might have caused death if it were more severe.

• Requires hospitalization or a prolongation of an existing hospitalization

In general, hospitalization signifies that the participant has been detained at the hospital or emergency department for observation or treatment that would not have been appropriate in the physician's office or outpatient setting. Complications that occur during hospitalization are AEs, but not necessarily SAEs. An occurrence or complication that prolongs hospitalization is an SAE. When there is doubt as to whether hospitalization occurred or was necessary, the AE should be considered an SAE. Hospitalization for elective treatments of a preexisting condition that did not worsen from its original baseline level is not considered an SAE.

 A persistent or significant incapacity or substantial disruption of the ability to conduct normal life functions

This definition is not intended to include AEs of relatively minor medical significance, such as uncomplicated headache, nausea, vomiting, diarrhea, influenza, or accidental trauma (e.g., sprained ankle) that may interfere or prevent everyday life functions but do not constitute a substantial disruption.

• A congenital anomaly or birth defect

# • Other important medical events

Medical or scientific judgment should be exercised in deciding whether reporting is appropriate for other important medical events that may not result in death, be life threatening, or require hospitalization but still may jeopardize the participant or may require medical intervention to prevent one of the outcomes listed in this definition. These events should also be considered serious. Examples of such events are intensive treatment in an emergency room or at home for allergic bronchospasm, blood dyscrasias, or convulsions that do not result in hospitalization, or development of drug dependency or drug abuse.

An SAE requires additional detailed reports and follow-up. The content of these detailed reports must address the investigator's estimate of causality. The medical monitor will review the SAE to determine if it is an expected SAE (i.e., whether or not the SAE is identified in nature, severity, or frequency in the Investigator's Brochure).

The investigator is responsible for performing periodic and specific assessments for SAEs at study visits. The investigator and clinical staff will note all SAEs mentioned by the participant during and after administration of the investigational product until the end of the study. All clinical complaints volunteered by, or elicited from, the participant during the study will be recorded on the appropriate page of the source documentation for the indicated study period. Information related to serious adverse events will be recorded on the eCRF. The participant will receive appropriate treatment guidance for any SAE that occurs.

All SAEs judged to be clinically significant, including clinically significant laboratory abnormalities, will be followed until resolution or considered stable by the investigator. All SAEs will be summarized in the annual report or more frequently, if requested by the regulatory agency. Serious adverse events require special reporting in addition to documentation in the eCRF as described in Section 6.2.

### 6.2 RECORDING SERIOUS ADVERSE EVENTS

When an SAE occurs, the investigator is responsible for reviewing all documentation (e.g., hospital progress notes, laboratory and diagnostic reports) relevant to the event(s). The investigator will record all relevant information about

the SAEs on the SAE page of the eCRF. It is not acceptable for the investigator to send photocopies of the participant's medical records in lieu of the properly completed SAE pages of the eCRF. These types of documents should not be sent unless they are specifically requested by pharmacovigilance. If this request occurs, all participant identifiers and protected health information will be blinded on the copies of the medical records before submission to the appropriate authorities.

The investigator will also attempt to report a diagnosis versus signs, symptoms, or other clinical information for the SAE. The diagnosis, not the individual signs and symptoms, should be documented on the appropriate page of the eCRF as the SAE. In addition, SAEs need to be reported on the SAE report form.

# 6.3 ASSESSMENT OF SEVERITY

The investigator will assess the severity for each SAE reported during the study. The assessment will be based on the investigator's clinical judgment.

The classifications in Table 2 should be used in assigning severity of each AE recorded in the eCRF. Additional guidance is provided in Appendix B for specific AEs, laboratory abnormalities, and changes in vital signs.

Table 2. Classification of AEs by Severity

| | <u> </u> |
|---|---|
| Severity | Definition |
| Grade 1<br>Mild AE | Transient or mild discomfort (<48 hours); no medical intervention or therapy required |
| Grade 2<br>Moderate AE | Mild to moderate limitation in activity, some assistance may be needed; no or minimal medical intervention or therapy required |
| Grade 3<br>Severe AE | Marked limitation in activity, some assistance usually required; medical intervention or therapy required, hospitalization possible |
| Grade 4 Life-threatening AE or Death | Extreme limitation in activity, significant assistance required; significant medical intervention or therapy required, hospitalization or hospice care probable |

AE = adverse event.

Any SAE that changes in severity during its course will be recorded in the eCRF at the highest level experienced by the participant.

Severity of an AE is graded as follows: Mild, moderate, severe or life-threatening myocardial infarction. An AE that is assessed as severe should not be confused with an SAE. An event may be of relatively minor medical significance, such as a severe headache, but not be considered an SAE. Both AEs and SAEs can be

assessed as severe. An AE is defined as serious when it meets one of the predefined outcomes as described in Section 6.1.

### 6.4 ASSESSMENT OF CAUSALITY

The investigator must estimate the relationship between the investigational product and the occurrence of each SAE by using his or her best clinical judgment. Elements to consider include the history of the underlying disease, concomitant therapy, other risk factors and the temporal relationship of the event to the investigational product. The investigator will also consult the Investigator's Brochure or product-labeling information for marketed products in estimating the relationship.

Because of reporting timelines, the investigator might have minimal information to include in the initial SAE report. However, the investigator must always make an assessment of causality for every event prior to the transmission of the SAE report. The investigator may change his or her opinion of the causality in light of follow-up information, with subsequent amendment of the SAE report. Causality assessment is one of the criteria used to determine regulatory reporting requirements and should not be left blank. Table 3 provides the definitions to use in the assessment.

CDPH rBV A/B

IND 015155

 Table 3.
 Assessment of Causality of Adverse Events

| Term | Definition |
|---|---|
| Definitely | The AE follows a reasonable temporal sequence from treatment and is consistent with the Investigator's Brochure. |
| Probably | <ul> <li>The AE follows a reasonable temporal sequence from the<br/>administration of the investigational drug.</li> </ul> |
| | • The AE cannot be easily explained from the participant's clinical condition, environmental or toxic factors, or other therapy administration. |
| | <ul> <li>The AE disappears or diminishes on cessation or reduction in<br/>dose, except in case of irreversible damage (positive de-<br/>challenge).</li> </ul> |
| | • The AE follows a known pattern or response of the investigational drug. |
| | The AE reappears upon re-administration of the investigational drug (positive re-challenge). |
| Possibly | <ul> <li>The AE follows a reasonable temporal sequence from the<br/>administration of the investigational drug.</li> </ul> |
| | <ul> <li>The AE cannot easily be explained from the participant's<br/>clinical condition, environmental or toxic factors, or other<br/>therapy administration.</li> </ul> |
| | <ul> <li>The AE follows a known pattern or response of the<br/>investigational drug.</li> </ul> |
| | <ul> <li>The AE disappears or diminishes on cessation or reduction in<br/>dose, except in case of irreversible damage (positive de-<br/>challenge).</li> </ul> |
| Unlikely | <ul> <li>The AE follows a reasonable temporal sequence from<br/>administration of the investigational drug.</li> </ul> |
| | <ul> <li>The AE can be easily explained from the participant's clinical<br/>condition, environmental or toxic factors, or other therapy<br/>administration.</li> </ul> |
| | The AE does not follow a known response pattern of the investigational drug. |
| Not Related | • The AE does not follow a reasonable temporal sequence from administration of the investigational drug and occurrence of the AE. |
| | <ul> <li>The AE could readily have been produced by the participant's<br/>clinical state, environmental or toxic factors, or other therapy<br/>administration.</li> </ul> |
| | <ul> <li>The AE does not follow a known response pattern to the<br/>investigational drug.</li> </ul> |
| | • The AE does not reappear or worsen when the investigational drug is re-administered (negative re-challenge). |

AE = adverse event.

### 6.5 EXPECTEDNESS OF ADVERSE EVENTS

An expected AE is one that is consistent with the known risk information described in the current Investigator's Brochure. An AE is considered unexpected if it is not listed the in the Investigator's Brochure or it is not listed at the specificity or severity that has been observed. This will be assessed by the medical monitor or sponsor-investigator upon receipt of the initial AE report.

#### 6.6 ADVERSE EVENTS OF SPECIAL INTEREST

Adverse events of special interest that are particularly specific to this study will be collected, assessed and recorded in the eCRF as an AE. These events of special interest will be collected in addition to the SAEs described in Section 6.1 and include the following clinical situations (see Section 3.3.2):

- Frequency of injection site reactions and systemic reactions among the study participants that are assessed as severe between Day 0 and 7 will be captured as an AE.
- Clinically significant changes in hematology between screening and Week 4 that are assessed as severe will be captured as an AE.

### 6.7 REPORTING OF SERIOUS ADVERSE EVENTS

Any SAE occurring after the participant has been vaccinated with rBV A/B must be reported to the medical monitor and sponsor-investigator by phone, fax, or email within 24 hours of the time the investigator becomes aware of the SAE (Table 4). Urgent reporting of SAEs is required for the following reasons:

- 1. To enable the sponsor-investigator to fulfill the reporting requirements to the appropriate regulatory authority
- 2. To facilitate the sponsor-investigator's rapid dissemination of information about SAEs to other investigators or sites in a multicenter study
- 3. To facilitate reporting unanticipated and/or serious problems involving risk to participants to the IRB within 48 hours.

CONFIDENTIAL **CDPH** rBV A/B

Clinical Protocol IND 015155

Table 4. Timeline for Reporting Serious Adverse Events to Medical Monitor and Sponsor-Investigator

| Initial SAE Report | | Follow-up SAE Report | |
|--------------------|------------|----------------------|--------------------|
| Time Frame | Documents | Time Frame | Documents |
| 24 hours | SAE report | 7 days | Updated SAE report |

SAE = serious adverse event.

The SAE report form will be completed as thoroughly as possible, including the following information:

- Participant identification information
- All available details about the event
- Causality of each SAE
- Signature of the investigator

The SAE report will be forwarded to the DSMB within the designated time frames. If the investigator does not have all information about an SAE, the investigator will NOT wait to receive additional information before notifying the DSMB of the SAE and completing the form. The form will be updated when additional information is received.

IND Safety Reports: The investigator will report a suspected adverse reaction that is both "serious" and "unexpected" to FDA in accordance with the timeframe outlined in 21 CFR 312.32. FDA and all participating investigators will be notified of potentially serious risks identified from any source within 15 calendar days after the sponsor-investigator receives the safety information and determines that it is reportable [21 CFR312.32 (c) (1)]. The sponsor-investigator must also notify FDA of any unexpected fatal or life-threatening suspected adverse reaction as soon as possible but in no case later than 7 calendar days after the sponsor-investigator's initial receipt of the information

### 6.8 FOLLOW-UP OF SERIOUS ADVERSE EVENTS

All SAEs (as well as clinically significant changes in hematology that result in a severe or serious adverse event) will be followed until the occurrence of one of the following:

- The event resolves.
- The condition stabilizes.
- The event is otherwise explained.
- The participant is lost to follow-up.

The appropriate SAE report form will be updated for SAEs only once the SAE resolves, stabilizes, is otherwise explained, or the participant is lost to follow-up. The investigator will also ensure that additional updates include any supplemental data that may explain causality of the event(s).

New or updated information will be recorded on a copy of the initially completed SAE report, with all the changes signed and dated by the investigator or designee. The updated SAE report will then be signed by the investigator and resubmitted to the DSMB as outlined in Table 4.

# 6.9 INJECTION SITE AND SYSTEMIC REACTIONS

Commonly seen injection site reactions for rBV A/B are consistent with reactions in participants vaccinated with other recombinant protein vaccines that include Alhydrogel<sup>™</sup>. The majority of reactions at the injection site seen to date with rBV A/B have been mild or moderate in severity and included erythema, pain, pruritus, and swelling. Participants will be actively monitored for localized and systemic reactions to the injections and an anaphylaxis (epinephrine) kit will be available at the time of injections.

The definitions to be used to determine severity of injection site reactions are provided in Table 5.

CONFIDENTIAL CDPH rBV A/B Clinical Protocol IND 015155

Table 5. Protocol Definitions for Severity of Injection Site, ie., Local Reactions

| Local Reaction<br>to Injectable<br>Product | Mild<br>(Grade 1) | Moderate<br>(Grade 2) | Severe<br>(Grade 3) | Potentially<br>Life-Threating<br>(Grade 4) |
|---|---|---|---|---|
| Injection site pain | Does not interfere with activity | Repeated use of<br>nonnarcotic<br>pain reliever<br>>24 hours or<br>interferes with<br>activity | Any use of narcotic pain reliever or prevents daily activity | ER visit or<br>hospitalization |
| Injection site tenderness | Mild discomfort<br>to touch | Discomfort with movement | Significant discomfort at rest | ER visit or hospitalization |
| Injection site<br>erythema<br>(redness) <sup>a</sup> | 2.5-5.0 cm | 5.1-10.0 cm | >10.0 cm | Bullae, necrosis,<br>or exfoliative<br>dermatitis |
| Injection site<br>swelling<br>(induration) <sup>b</sup> | 2.5-5.0 cm and does not interfere with activity | 5.1-10.0 cm or interferes with activity | >10.0 cm or<br>prevents daily<br>activity | Necrosis |

ER = emergency room.

Systemic reactions collected in the diary are severity of muscle weakness, malaise, rash, headache, nausea, chest discomfort, breathing difficulties, anxiety, feelings of depression, and neuromuscular TEAEs. For systemic reactions, use the guidance provided in Appendix B.

### 6.10 DATA AND SAFETY MONITORING BOARD

The DSMB will meet quarterly throughout the study and as needed as described in Section 4.4. The specific information that will be reviewed to make its recommendation will be safety data and neutralizing antibody concentrations.

In addition, the DSMB will convene at any time during the study if a stopping rule is met (see Section 4.4.2)

# 6.11 PREGNANCY

If a participant becomes pregnant at any time after receipt of the study vaccine, she should report the pregnancy via telephone to the study investigators within 24 hours

In addition to grading the measured local reaction at the greatest single diameter, the measurement should be recorded as a continuous variable.

Induration (swelling) should be evaluated and graded using the functional scale as well as the actual measurement.

rBV A/B
Clinical Protocol IND 015155

of being made aware of it; study investigators will then promptly complete the pregnancy report form and forward the form to the medical monitor and sponsor-investigator. The female participant will be discontinued from further study procedures, including plasmapheresis. The pregnancy will be followed until there is an outcome and the outcome is reported to the study investigators.

# 7.0 STUDY OR SITE TERMINATION AND PARTICIPANTDISCONTINUATION

### 7.1 PARTICIPANT DISCONTINUATION

Participants will be encouraged to complete the study; however, they may voluntarily withdraw at any time. The investigator will provide a written explanation of the reason for discontinuation in a source document, which will be transcribed to the appropriate eCRF page. If a participant withdraws before completion, every effort should be made to complete the assessments scheduled during the final on-site study visit. In addition, the participant will be offered safety follow-up for the planned duration of the study (through the Week 26 telephone contact) regardless of the reason for discontinuation.

A participant may be removed from the study for the reasons described in Section 7.1.1 through Section 7.1.5.

### 7.1.1 Adverse Event

If a participant suffers an AE that, in the judgment of the investigator, the sponsor-investigator, or the medical monitor, presents an unacceptable consequence or risk to the participant, the participant may be discontinued from the study.

# 7.1.2 Intercurrent Illness

A participant may be discontinued from the study if, in the judgment of the investigator, the participant develops an intercurrent illness or complication that is not consistent with the protocol requirements or that, in any way, justifies withdrawal from the study.

# 7.1.3 Noncompliance

After consultation among the investigator, the medical monitor, and study/data monitor, a participant may be discontinued from the study for failure to comply with protocol requirements. Upon being discontinued from the study, the participant will be notified by study personnel and the reason for discontinuation documented in the appropriate eCRF page and on study source documents.

# 7.1.4 Refusal of Investigational Product Administration

Any participant refusing vaccination with rBV A/B for any reason will be discontinued from the study, and the reason(s) will be documented on the appropriate eCRF page. Efforts should be made to monitor the participant for AEs and to complete follow-up assessments after discontinuation. These efforts should be documented on the appropriate eCRF page.

# 7.1.5 Withdrawal of Consent

Any participant that withdraws consent for any reason at any time during the study will be discontinued from the study, and the reason(s) will be documented on the appropriate eCRF page.

### 7.2 PREMATURE STUDY OR SITE TERMINATION

If the sponsor, investigator, medical monitor, study/data monitor, or appropriate regulatory officials discover conditions arising during the study that indicate that the study should be halted or that the site should be terminated, this action may be taken after appropriate consultation among the sponsor-investigator, medical monitor, and study/data monitor. Conditions that may warrant termination of the study include, but are not limited to, the following:

- The discovery of an unexpected, serious, or unacceptable risk to the participants enrolled in the study
- A decision on the part of the sponsor-investigator or product manufacturer to suspend or discontinue testing, evaluation, or development of the product

A study conducted at a single site in a multicenter study may also warrant termination under the following conditions:

- Failure of the investigator to enroll participants into the study at an acceptable rate
- Failure of the investigator to comply with pertinent regulations of appropriate regulatory authorities

CONFIDENTIAL **CDPH** rBV A/B

Clinical Protocol IND 015155

> Submission of knowingly false information from the site to the sponsor-investigator, study/data monitor, or appropriate regulatory authority

Insufficient adherence to protocol requirements

Study termination and follow-up will comply with the conditions set forth in the ICH E6 Guideline for Good Clinical Practice, Sections 4.12, 4.13, 5.20, and 5.21.

# 8.0 DATA COLLECTION AND PROCESSING AND STATISTICAL ANALYSIS

### 8.1 DATA COLLECTION AND PROCESSING

eCRFs will be used to capture study assessments and data. The study investigator or other delegated study personnel will enter data from source documents into the eCRFs. All eCRFs and their data will be reviewed and source verified by the study/data monitor. The medical monitor may examine the eCRFs for preliminary medical review. Once the eCRFs are completed and source-verified, the study investigator will sign and date all required pages, thereby verifying the accuracy of all data contained in the eCRFs.

# 8.2 STATISTICAL ANALYSIS

### **8.2.1** General Overview

The data will be summarized in tables listing the mean, standard deviation or standard error, median, minimum, maximum and number of participants for continuous data or in tables listing count and percentage for categorical data, where appropriate. Data will be listed by "participant ID." All statistical analyses will be performed and data appendices will be created by using SAS.

# **8.2.2** Populations of Interest

# **8.2.2.1** Immunogenicity Population

The immunogenicity population defines participants who have received the vaccine dose, have a baseline NAC, and have at least one post-vaccination immunogenicity assessment up to and including 4 weeks after administration of rBV A/B.

# **8.2.2.2** Per Protocol Population

The per protocol population defines participants who have received the vaccine dose, have a baseline NAC, and have the relevant immunogenicity assessments completed within the protocol-specified timelines (including visit windows) for the time point(s) summarized and who do not have major protocol violations expected to affect immunogenicity. Determination of a major protocol violation expected to

affect immunogenicity will be done by the sponsor-investigator before reviewing the immunogenicity data for the applicable participant. The precise reasons for excluding participants from the per protocol population will be fully defined and documented. (Note: It is possible for a participant to be included in the primary per protocol analysis for Week 4, even if the subsequent blood draws occur outside of the study windows.)

# 8.2.2.3 Safety Population

The safety population comprises all participants enrolled into the study who received the vaccine dose and had at least one post-baseline safety assessment (this assessment can include a response from a participant that no adverse events occurred).

# 8.2.2.4 Plasma-Donating Population

The plasma-donating population will include all participants who receive the vaccine and donate at least one plasma unit.

# 8.2.3 Baseline Comparability

No formal baseline comparability testing is planned for this study.

# 8.2.4 Immunogenicity Analysis

The immunogenicity population will be used for all immunogenicity endpoints. The per protocol population will be used in the case that any sensitivity analyses are deemed necessary.

The immunogenicity parameters are concentrations of neutralizing antibodies against botulinum toxin type A and toxin type B. These parameters will be analyzed by using NAC data from a validated mouse neutralization assay.

For the primary endpoint, a positive response will be defined as achieving a greater than or equal to four times increase (point estimate) above baseline in NAC by Week 4 compared with Week 0 in at least 50% of the participants in the immunogenicity population for botulinum toxin type A and type B, respectively.

A point estimate and two-sided 95% confidence interval for the proportion of participants who achieve this endpoint will be provided.

For the first secondary immunogenicity endpoint, a positive response will be defined as achieving a two times increase above baseline in the estimated area under the plasma NAC-time curve in the period from Week 0 to Week 12 in comparison to straight-line extension of the Week 0 antibody concentration from Week 0 to Week 12 in least 50% of the participants.

For the second secondary immunogenicity endpoint, a positive response will be defined as is achieving a three times or greater increase in NAC above baseline by Week 4 in at least 50% of the participants for botulinum toxin type A and type B. A point estimate and two-sided 95% confidence interval for the proportion of participants who achieve this endpoint will be provided.

Further details of the analysis, will be provided as needed in a separate statistical analysis plan.

In the event that the primary endpoint is not met for neutralizing antibodies against botulinum toxin type A and type B, the sponsor-investigator will determine if the plasma collected during the study contains sufficient antibody titers for meeting specifications for BabyBIG production. If the immune responses meet specifications to permit the production of BabyBIG, then the trial will still be considered successful. Also, a second booster dose of rBV A/B vaccine may be considered; however, this will require operational modifications (e.g., a protocol amendment and updated consent form).

# 8.2.5 Safety Analysis

The safety analysis will use the safety population.

Localized and systemic severe AEs and SAEs collected from the Week 1 telephone call will be summarized by category and severity. A point estimate of incidence, with 95% confidence limits will be computed and reported (not coded into the Medical Dictionary for Regulatory Activities [MedDRA] terminology or assessed for relatedness). The time period summarized will include throughout the study as a whole and again within Days 0 through 7. For tables summarizing severity, the

highest reported severity grade will be used. In addition, the average duration, by category, will be summarized.

All other SAE data will be listed individually and summarized by system organ class and preferred terms for each treatment group. When calculating the incidence of SAEs, each SAE based on preferred terminology from MedDRA will be counted only once for a given participant. If the same SAE occurs on multiple occasions in a participant, the occurrence with the highest severity and highest causality relationship to the vaccine will be reported. If two or more SAEs are reported as a unit, the individual terms will be reported as separate experiences.

Treatment-emergent abnormal values that occur prior to the end of the study will be summarized. Laboratory abnormalities will be assessed for relatedness. Treatment-emergent changes from normal to abnormal values in key laboratory parameters will be identified.

Presentation of relatedness in tables will be based on the investigator's assessment.

# 8.2.6 Sample Size

No formal power calculations will be performed for this study. The sample size will consist of up to 50 participants. On the basis of prior sponsor-investigator experience, this sample size is considered adequate for fulfilling the study objectives.

### 9.0 CLINICAL STUDY ADMINISTRATION

# 9.1 INFORMED CONSENT WITH AUTHORIZATION FOR USE AND DISCLOSURE OF PROTECTED HEALTH INFORMATION

Written informed consent with authorization of use and disclosure of protected health information must be obtained from each participant before performing any study-specific screening/baseline period evaluations. The informed consent form that includes authorization for use and disclosure of protected health information must have been reviewed and approved by the sponsor-investigator, the study/data monitor, and the investigator's IRB prior to the initiation of the study. The ICF will conform to the 20 elements of informed consent described in ICH E6, Section 4.8 and will include the elements required by Title 45 of the Code of Federal Regulations, Section 164.508(b) and any local regulations for valid authorizations. One copy of the signed ICF with authorization for use and disclosure of protected health information form will be given to the participant, and the investigator will retain the original in the Investigators' Study Files.

### 9.2 STUDY DOCUMENTATION

# 9.2.1 Investigator Information

Investigator information is included in the study procedure manual, which is updated as needed.

# 9.2.2 Investigators' Study Files

Documentation about the investigator and study staff, the IRB, and the institution is required before study site initiation. Copies of these documents will be kept on-site in study site—specific binders or files, along with the following supplemental information: a list of investigator's obligations; the current Investigator's Brochure; the clinical trial protocol and amendments; safety information; information about investigational product, biological samples, and the laboratory; the study procedure manual and study logs; and records of monitoring activities.

The investigator is responsible for ensuring frequent backup of all electronic data systems used for primary documentation or source documentation. Electronic

(eCRF) data will be backed up periodically as described in the EDC vendor's standard operating procedures.

# 9.2.3 Case Report Forms and Source Documentation

The investigator must make study data accessible to the study/data monitor, other authorized representatives of the sponsor-investigator, and the appropriate regulatory authority inspectors. The eCRF for each participant will be checked against source documents at the study site by the study/data monitor, and a final copy of the eCRF will be signed by the investigator with an electronic signature. A copy of the final eCRFs will be provided to the investigator in portable document format on computer disc after study closure to be kept in the investigator's study files.

# 9.2.4 Retention of Study Documents

According to ICH E6, Section 4.9, all eCRFs, as well as supporting paper and electronic source documentation and administrative records, must be retained by the investigator until at least 2 years after the last approval of a marketing application and until there are no pending or contemplated marketing applications or until at least 2 years have elapsed since the formal discontinuation of clinical development of the investigational product in the United States. The sponsor-investigator is responsible for informing the investigator and institution as to when these documents no longer need to be retained. No study documents will be destroyed or moved to a new location without prior written approval from the sponsor-investigator. If the investigator relocates, retires, or withdraws from the clinical study for any reason, all records required to be maintained for the study should be transferred to a designee approved by the sponsor-investigator, such as another investigator at the institution where the study was conducted.

Audit trails for electronic documents must be retained for a period at least as long as that required for the participant electronic records to which they pertain. The investigator must retain either the original or a certified copy of audit trails.

CONFIDENTIAL CDPH rBV A/B Clinical Protocol IND 015155

# 9.3 CONFIDENTIALITY

### 9.3.1 Data

The investigator shall keep all information about the nature of the proposed investigation provided by the sponsor-investigator or study monitor to the investigator confidential (with the exception of information required by law or regulations to be disclosed to the IRB, the participant, or the appropriate regulatory authority). Additionally, de-identified data (safety and immunological) will be disclosed to DynPort Vaccine Company LLC to be used for safety reporting required by regulatory authorities.

# 9.3.2 Participant Anonymity

The anonymity of participating participants must be maintained. Participants will be identified by an assigned participant number on eCRFs and other documents retrieved from the site or sent to the study/data monitor, sponsor-investigator, regulatory agencies, central laboratories, or blinded reviewers. Documents that identify the participant (e.g., the signed informed consent form) must be maintained in strict confidence by the investigator and designated study staff, except to the extent necessary to allow auditing by the appropriate regulatory authority, the study/data monitor, or sponsor-investigator representatives.

### 9.4 PROTOCOL COMPLIANCE AND AMENDMENT PROCEDURES

Substantive changes in the protocol include changes that affect the safety of participants or changes that meaningfully alter the scope of the investigation, the scientific quality of the study, the experimental design, dosages, assessment variable(s), the number of participants treated, or the participant selection criteria. Such changes must be prepared as a protocol amendment by the sponsor-investigator and implemented only upon joint approval of the sponsor-investigator and the IRB. In parallel with the IRB approval process, the protocol amendment will be submitted to the appropriate regulatory authority as an amendment to the regulatory submission under which the study is being conducted. If a protocol amendment requires changes in the informed consent form, the revised informed consent form prepared by the investigator must also be approved by the sponsor-investigator, study/data monitor, and the IRB before implementation.

rBV A/B
Clinical Protocol IND 015155

Deviations from the protocol are allowed only in situations for which the deviation would eliminate an immediate risk to a participant and that are deemed crucial for the safety and well-being of that participant. The investigator or the attending physician also will contact the medical monitor as soon as possible in the case of such a deviation. These deviations do not require preapproval by the IRB; however, the IRB and medical monitor must be notified in writing or via e-mail as soon as possible after the deviation occurs. In addition, the investigator will document in the participant's eCRF the reasons for the protocol deviation and the ensuing events.

# 9.5 STUDY/DATA MONITOR FUNCTIONS AND RESPONSIBILITY

The study/data monitor, in accordance with the sponsor-investigator's requirements, will ensure that the clinical trial is conducted and documented properly by carrying out the activities outlined in ICH E6, Section 5.18.4.

rBV A/B
Clinical Protocol IND 015155

# 10.0 REFERENCES

1. Centers for Disease Control and Prevention. Notice of CDC's discontinuation of investigational pentavalent (ABCDE) botulinum toxoid vaccine for workers at risk for occupational exposure to botulinum toxins. MMWR 2011;60(42):1454-1455.

2. U.S. Department of Health and Human Services, Food and Drug Administration. Code of Federal Regulations Title 21, Part 640 additional standards for human blood and blood products. Revised 01 April 2013; Available at:

http://www.accessdata.fda.gov/scripts/cdrh/cfdocs/cfcfr/CFRSearch.cfm? CFRPart=640&showFR=1&subpartNode=21:7.0.1.1.7.7.

CONFIDENTIAL CDPH rBV A/B Clinical Protocol IND 015155

# **APPENDICES**

rBV A/B
Clinical Protocol IND 015155

# **APPENDIX A**

# CODE OF FEDERAL REGULATIONS PART 640: ADDITIONAL STANDARDS FOR HUMAN BLOOD AND BLOOD PRODUCTS

# CODE OF FEDERAL REGULATIONS PART 640—ADDITIONAL STANDARDS FOR HUMAN BLOOD AND BLOOD PRODUCTS

Subpart G—Source Plasma

§ 640.63 Suitability of donor.

- (a) *Method of determining*. The suitability of a donor for Source Plasma will be determined by a qualified licensed physician or by persons under his or her supervision and trained in determining donor suitability. Such determination will be made on the day of collection from the donor by means of a medical history, tests, and such physical examination as appears necessary to the qualified licensed physician.
- (b) Initial medical examinations.
  - (1) Each donor will be examined by a qualified licensed physician on the day of the first donation or no more than 1 week before the first donation and at subsequent intervals of no longer than 1 year.

(2)

- (i) A donor who is to be immunized for the production of high-titer plasma will be examined by a qualified licensed physician. The medical examination will be performed within no more than 1 week before the first immunization injection. The medical examination for plasmapheresis need not be repeated, if the first donation occurs within 3 weeks after the first injection.
- (ii) A donor who is an active participant in a plasmapheresis program, and has been examined in accordance with paragraph (b)(1) of this section, need not be reexamined before immunization for the production of high-titer plasma.
- (3) Each donor will be certified to be in good health by the examining physician. The certification of good health will be on a form supplied by the licensed establishment and will indicate that the certification applies to the suitability of the individual to be a plasmapheresis donor and, when applicable, an immunized donor.

Clinical Protocol

- indicated in part by:
- (1) Normal temperature;

(c)

(2) Demonstration that systolic and diastolic blood pressures are within normal limits, unless the examining physician is satisfied that an individual with blood pressures outside these limits is an otherwise qualified donor under the provisions of this section;

Qualification of donor. Donors will be in good health on the day of donation, as

- (3) For female donors, a blood hemoglobin level of no less than 12.5 g of hemoglobin per 100 mL of blood or a hematocrit level of 38% (female donors may have a hemoglobin level of between 12.0 and 12.5 g hemoglobin per 100 mL of blood, or a hematocrit between 36 and 38% provided additional steps ensure the health of the donor will not be adversely affected due to donation); For male donors, a blood hemoglobin level of no less than 13.0 g of hemoglobin per 100 mL, or a hematocrit level no less than 39%;
- (4) A normal pulse rate;
- (5) A total serum or total plasma protein of no less than 6.0 g per 100 mL of blood;
- (6) Weight, which will be at least 110 pounds;
- (7) Freedom from acute respiratory diseases;
- (8) Freedom from any infectious skin disease at the site of phlebotomy and from any such disease generalized to such an extent as to create a risk of contamination of the plasma;
- (9) Freedom from any disease, other than malaria, transmissible by blood transfusion, insofar as can be determined by history and examinations indicated in this section;
- (10) Freedom of the arms and forearms from skin punctures or scars indicative of addiction to self-injected narcotics;
- (11) Freedom from a history of viral hepatitis after the 11th birthday;
- (12) Freedom from a history of close contact within 12 months of donation with an individual having viral hepatitis;
- (13) Freedom from a history of having received, within 12 months, human blood or any derivative of human blood that the Food and Drug Administration has advised the blood establishment is a possible source of viral hepatitis, except for specific immunization performed in accordance with 640.66.

CDPH rBV A/B

IND 015155

CONFIDENTIAL **CDPH** rBV A/B IND 015155

Clinical Protocol

General. Any donor who, in the opinion of the interviewer, appears to be under the (d) influence of any drug, alcohol, or for any reason does not appear to be providing reliable answers to medical history questions, will not be considered a suitable donor.

- (e) Failure to return red blood cells. Any donor who has not had the red blood cells returned from a unit of blood collected during a plasmapheresis procedure or who has been a donor of a unit of whole blood will not be subjected to plasmapheresis for a period of 8 weeks, unless:
  - (1) The donor has been examined by a qualified licensed physician and certified by the physician to be acceptable for further plasmapheresis before expiration of the 8-week period;
  - (2) The donor possesses an antibody that is
    - (i) transitory,
    - (ii) of a highly unusual or infrequent specificity, or
    - (iii) of an unusually high titer; and
  - (3) The special characteristics of the antibody and the need for plasmapheresing the donor are documented.

rBV A/B
Clinical Protocol IND 015155

# **APPENDIX B**

TOXICITY TABLES FROM GUIDANCE FOR INDUSTRY: TOXICITY GRADING SCALE FOR HEALTHY ADULT AND ADOLESCENT PARTICIPANTS ENROLLED IN PREVENTIVE VACCINE CLINICAL TRIALS

rBV A/B Clinical Protocol IND 015155

| Vital Signs <sup>a</sup> | Mild<br>(Grade 1) | Moderate<br>(Grade 2) | Severe<br>(Grade 3) | Potentially Life<br>Threatening<br>(Grade 4) |
|---|---|---|---|---|
| Fever (°C) <sup>b</sup> | 38.0-38.4 | 38.5-38.9 | 39.0-40.0 | >40.0 |
| (°F) <sup>b</sup> | 100.4-101.1 | 101.2-102.0 | 102.1-104.0 | >104.0 |
| Tachycardia<br>(beats per minute) | 101-115 | 116-130 | >130 | ER visit or<br>hospitalization fo<br>arrhythmia |
| Bradycardia <sup>c</sup> (beats per minute) | 50-54 | 45-49 | <45 | ER visit or<br>hospitalization fo<br>arrhythmia |
| Hypertension: systolic<br>(mm Hg) | 141-150 | 151-155 | >155 | ER visit or<br>hospitalization for<br>malignant<br>hypertension |
| Hypertension: diastolic<br>(mm Hg) | 91-95 | 96-100 | >100 | ER visit or<br>hospitalization for<br>malignant<br>hypertension |
| Hypotension: systolic<br>(mm Hg) | 85-89 | 80-84 | <80 | ER visit or<br>hospitalization for<br>hypotensive shoo |
| Respiratory rate (breaths per minute) | 17-20 | 21-25 | >25 | Intubation |

 $\overline{ER}$  = emergency room.

CDPH

a Participant should be at rest for all vital sign measurements.

Oral temperature should be taken, and there should be no consumption of recent hot or cold beverages or smoking.

c Use clinical judgment when characterizing bradycardia among some healthy participant populations, for example conditioned athletes.

Table 7. Systemic Clinical Abnormalities

| Systemic<br>(General) | Mild<br>(Grade 1) | Moderate<br>(Grade 2) | Severe<br>(Grade 3) | Potentially Life<br>Threatening<br>(Grade 4) |
|---|---|---|---|---|
| Nausea/vomiting | No interference<br>with activity, or 1<br>to 2 episodes per<br>24 hours | Some interference<br>with activity or<br>>2 episodes per<br>24 hours | Prevents daily<br>activity, requires<br>outpatient<br>intravenous<br>hydration | ER visit or<br>hospitalization for<br>hypotensive shock |
| Diarrhea | 2 to 3 loose stools<br>or <400 g per<br>24 hours | 4 to 5 stools or<br>400 to 800 g per<br>24 hours | 6 or more watery<br>stools or >800 g<br>per 24 hours or<br>requires outpatient<br>intravenous<br>hydration | ER visit or<br>hospitalization |
| Headache | No interference with activity | Repeated use of<br>nonnarcotic pain<br>reliever >24 hours<br>or some<br>interference with<br>activity | Significant; any use of narcotic pain reliever or prevents daily activity | ER visit or hospitalization |
| Fatigue | No interference with activity | Some interference with activity | Significant;<br>prevents daily<br>activity | ER visit or hospitalization |
| Myalgia | No interference with activity | Some interference with activity | Significant;<br>prevents daily<br>activity | ER visit or hospitalization |
| Illness or clinical<br>adverse event | No interference with activity | Some interference<br>with activity, but<br>not requiring<br>medical<br>intervention | Prevents daily<br>activity and<br>requires medical<br>intervention | ER visit or<br>hospitalization |

 $\overline{ER}$  = emergency room.

Clinical Protocol

| Seruma | Mild<br>(Grade 1) | Moderate<br>(Grade 2) | Severe<br>(Grade 3) | Potentially Life<br>Threatening<br>(Grade 4) <sup>b</sup> |
|---|---|---|---|---|
| Glucose: | 65–69 | 55–64 | 45–54 | <45 |
| hypoglycemia (mg/dL) | | | | |
| Glucose: | | | | Insulin |
| hyperglycemia fasting | | | | requirements o |
| (mg/dL); | 100-110 | 111–125 | >125 | hyperosmolar |
| random (mg/dL) | 110–125 | 126–200 | >200 | coma |
| Blood urea nitrogen (mg/dL) | 23–26 | 27–31 | >31 | Requires dialysis |
| Creatinine (mg/dL) | 1.5–1.7 | 1.8–2.0 | 2.1–2.5 | >2.5 or require dialysis |
| Alkaline phosphate: increase by factor | 1.1–2.0 × ULN | 2.1–3.0 × ULN | 3.1–10 × ULN | >10 × ULN |
| Liver function tests: ALT, AST, increase by factor | 1.1–2.5 × ULN | 2.6–5.0 × ULN | 5.1–10 × ULN | >10 × ULN |
| Bilirubin: when accompanied by any increase in liver function test, increase by factor | 1.1–1.25 × ULN | 1.26–1.5 × ULN | 1.51–1.75 × ULN | >1.75 × ULN |
| Bilirubin: when liver function test is normal, increase by factor | 1.1–1.5 × ULN | 1.6–2.0 × ULN | 2.0–3.0 × ULN | >3.0 × ULN |
| Potassium -<br>Hyperkalemia<br>(mEq/L) | 5.1–5.2 | 5.3–5.4 | 5.5–5.6 | >5.6 |
| Potassium -<br>Hypokalemia (mEq/L) | 3.5–3.6 | 3.3–3.4 | 3.1–3.2 | <3.1 |
| Calcium -<br>Hypocalcemia<br>(mg/dL) | 8.0–8.4 | 7.5–7.9 | 7.0–7.4 | <7.0 |
| Calcium -<br>Hypercalcemia<br>(mg/dL) | 10.5–11.0 | 11.1–11.5 | 11.6–12.0 | >12.0 |

ALT = alanine aminotransferase; AST = aspartate aminotransferase; ULN = upper limit of the normal range.

- The laboratory values provided in the table serve as guidelines and are dependent on institutional normal parameters. Institutional normal reference ranges should be provided to demonstrate that the laboratory values are appropriate.
- The clinical signs or symptoms associated with laboratory abnormalities might result in characterization of the laboratory abnormalities as potentially life-threatening (Grade 4). For example, a low potassium value that falls within a Grade 3 parameter should be recorded as a Grade 4 hypokalemia event if the participant had a new arrhythmia event associated with the low potassium value.

**Modified Hematology Clinical Abnormalities** Table 9.

| <b>Hematology</b> <sup>a</sup> | Mild<br>(Grade 1) | Moderate<br>(Grade 2) | Severe<br>(Grade 3) | Potentially Life<br>Threatening<br>(Grade 4) |
|---|---|---|---|---|
| Hemoglobin: female (g/dL) | 11.0-12.0 | 9.5-10.9 | 8.0-9.4 | <8.0 |
| Hemoglobin: male (g/dL) | 12.5-13.5 | 10.5-12.4 | 8.5-10.4 | <8.5 |
| WBC increase (cell/mm <sup>3</sup> ) | 10.800-15,000 | 15,001-20,000 | 20,001-25,000 | >25,000 |
| WBC decrease (cell/mm <sup>3</sup> ) | 2,500-3, 500 | 1,500-2,499 | 1,000-1,499 | <1,000 |
| Lymphocytes decrease (cell/mm³) | 750-1,000 | 500-749 | 250-499 | <250 |
| Neutrophils decrease (cell/mm <sup>3</sup> ) | 1,500-2,000 | 1,000-1,499 | 500-999 | <500 |
| Eosinophils (cell/mm <sup>3</sup> ) | 650-1,500 | 1,501-5,000 | >5,000 | Hypereosinophilic |
| Platelets decrease (cell/mm³) | 125,000-140,000 | 100,000-124,999 | 25,000-99,999 | <25,000 |

WBC = white blood count.

Table 10. **Clinical Abnormalities from Urinalysis Values** 

| | | | | Potentially Life |
|---|---|---|---|---|
| | Mild | Moderate | Severe | Threatening |
| Urine <sup>a</sup> | (Grade 1) | (Grade 2) | (Grade 3) | (Grade 4) |
| Protein | Trace | 1+ | 2+ | Hospitalization or |
| | | | | dialysis |
| Glucose | Trace | 1+ | 2+ | Hospitalization for |
| | | | | hyperglycemia |
| Blood (microscopic): | 1-10 | 11-50 | >50 and/or gross | Hospitalization or |
| red blood cells per | | | blood | packed red blood |
| high-power field | | | | cells transfusion |

The laboratory values provide in the table serve as guidelines and are dependent on institutional normal parameters. Institutional normal reference ranges should be provided to demonstrate that the laboratory values are appropriate.

The laboratory values provided in the table serve as guidelines and are dependent on institutional normal parameters. Institutional normal reference ranges should be provided to demonstrate that the laboratory values are appropriate.

**Table 11. Neuromuscular Toxicities** 

| | | | | Potentially<br>Life |
|---|---|---|---|---|
| Neurological Event | Mild<br>Grade 1 | Moderate<br>Grade 2 | Severe<br>Grade 3 | Threatening<br>Grade 4 |
| Muscle Weakness <sup>a</sup> | subjective<br>weakness with no<br>objective<br>symptoms or signs | mild objective<br>signs or<br>symptoms and<br>no decrease in<br>function | objective<br>weakness<br>function limited | paralysis |
| Ophthalmoplegia / Diplopia (double vision) | Intermittently<br>symptomatic,<br>intervention not<br>indicated | Symptomatic<br>and interfering<br>with function<br>but not with<br>interfering with<br>ADL; mild<br>objective signs<br>or symptoms;<br>intervention not<br>indicated | Symptomatic<br>and interfering<br>with function<br>and ADL;<br>objective<br>weakness;<br>medical<br>intervention<br>indicated | Disabling;<br>Paralysis;<br>medical<br>intervention<br>indicated |
| Vision – blurred vision<br>Vision - photophobia | Intermittently<br>symptomatic,<br>intervention not<br>indicated | Symptomatic<br>and interfering<br>with function<br>but not<br>interfering with<br>ADL; mild<br>objective signs<br>or symptoms | Symptomatic<br>and interfering<br>with function<br>and ADL;<br>objective<br>weakness; | Disabling |
| Voice changes / dysarthria<br>(e.g., hoarseness, loss or<br>alteration of voice) | Mild or<br>Intermittent<br>hoarseness or voice<br>change, but fully<br>understandable | Moderate or<br>persistent voice<br>changes, may<br>require<br>occasional<br>repetition but<br>understandable<br>on telephone | Severe voice<br>changes<br>including<br>predominantly<br>whispered<br>speech; may<br>require frequent<br>repetition or<br>face-to-face<br>contact for<br>understandability | Disabling; non-<br>understandable<br>voice or<br>aphonic; |
| Dyspnea<br>(shortness of breath) | Dyspnea on<br>exertion, but can<br>walk one flight of<br>stairs without<br>stopping | Dyspnea on<br>exertion, but<br>unable to walk<br>one flight of<br>stairs without<br>stopping | Dyspnea<br>interfering with<br>ADL | Dyspnea at rest; intubation may be indicated |
| Neuro-Cerebellar<br>(lack of coordination, tremor) | slight<br>incoordination<br>dysdiadochokinesis | intention<br>tremor,<br>dysmetria,<br>slurred speech;<br>nystagmus | locomotor ataxia | incapacitated |
| Cranial neuropathy | Asymptomatic, detected on examination | Symptomatic,<br>not interfering<br>with ADL | Symptomatic, interfering with ADL | Life-<br>threatening,<br>disabling |

<sup>&</sup>lt;sup>a</sup> Check for generalized, cranial muscles (see sentence below), extremities (upper and lower), and specific areas (extra ocular, facial, ocular, and trunk). Symptoms or signs of cranial muscle involvement are disruption of the appearance or functioning of the senses, facial muscles, pharynx, larynx, and neck.

CONFIDENTIAL CDPH rBV A/B Clinical Protocol IND 015155

# APPENDIX C PARTICIPANT DIARY

# Tolerability and Immunogenicity of a Single 40-µg Dose of Recombinant Botulinum Vaccine A/B (rBV A/B) for the Production of BabyBIG® in Volunteers with Existing Botulinum Immunity

# **Reaction Recording Sheet – Participant Home Diary**

| Study Site/Location*: | _/ | | | | | Parti | cipan | t Stud | dy ID | Numb | er*: _ | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Participant Name: | | | | | | | | | | | | | | |
| Recombinant vaccine given: | Date | : | | <u>/</u> | | | | _ Tim | ie: | | | | AM | / PM |
| | 1 d<br>24 | | 2 da<br>48 l | • | 3 da<br>72 h | | 4 da<br><u>96 h</u> | | 5 da<br>120 | | 6 da | - | 7 da<br>168 | - |
| Local reactions: | | | | | | | | | | | | | | |
| Soreness? | Υ | N | Y | N | Υ | N | Υ | N | Υ | N | Υ | N | Υ | N |
| Itching? | Υ | N | Υ | N | Υ | N | Υ | N | Υ | N | Υ | N | Υ | N |
| Erythema? (mm) <sup>a</sup> | | | | | | | | | | | | | | |
| Induration? (mm) <sup>a</sup> | | | | | | | | | | | | | | |
| Systemic reactions: | | | | | | | | | | | | | | |
| General malaise? | Υ | N | Υ | N | Υ | N | Υ | N | Υ | N | Υ | N | Υ | N |
| Fatigue? | Υ | N | Υ | N | Υ | N | Υ | N | Υ | N | Υ | N | Υ | N |
| Lethargy? | Υ | N | Υ | N | Υ | N | Υ | N | Υ | N | Υ | N | Υ | N |
| Chills, fever? | Υ | N | Υ | N | Υ | N | Υ | N | Υ | N | Υ | N | Υ | N |
| Lumps, soreness? (not local) | Υ | N | Y | N | Υ | N | Υ | N | Υ | N | Υ | N | Υ | N |
| Stiff back, stiff neck? | Υ | N | Υ | N | Υ | N | Υ | N | Υ | N | Υ | N | Υ | N |
| Nausea, vomiting, or diarrhea? | Υ | N | Y | N | Υ | Ν | Υ | N | Υ | N | Υ | Ν | Υ | N |
| Other GI symptoms? | Υ | N | Υ | N | Υ | N | Υ | N | Υ | N | Υ | N | Υ | N |
| Itching, hives? | Υ | N | Υ | N | Υ | N | Y | N | Υ | Ν | Υ | Ν | Υ | N |
| a Please use tool provided to me above: | easur | e. P | lease | list a | any n | nedic | ations | s use | d to t | reat t | he po<br>_ | tentia | l reac | tions |
| If you answered <b>yes</b> to any of the date/time of reaction, symptoms | abo | ve p | otent | ial rea | action | ns, ple | ease | recor | d add | itiona | –<br>I comi | ments<br>- | i.e., | |

If additional space required, please continue on back of this form.

Ver. August 2018

<sup>\*</sup> To be filled in by study staff

# APPENDIX D DONOR HISTORY QUESTIONNAIRE

# **PPTA Abbreviated Donor History Questionnaire For Frequent Plasma Donors**

This document is one component of the PPTA donor history questionnaire documents to be used by source plasma organizations. The PPTA abbreviated donor history questionnaire documents must be used collectively.





# PPTA Abbreviated Donor History Questionnaire For Frequent Plasma Donors

| Please Read the Medication List 2. Since you last donated plasma have you taken any medications on the medication list? Changes in Health Since you last donated plasma: Yes No 3. Female Donors: Have you been pregnant or are you pregnant now? 4. Have you had any new medical problems or diagnoses? 5. Have you had any new medical treatments, vaccinations or medications? 6. Have you had contact with someone who had a smallpox vaccination? 7. Have you donated whole blood, platelets or plasma at another center? Risk Activities Please review our Risk Poster Yes No |
|---|
| 2. Since you last donated plasma have you taken any medications on the medication list? Changes in Health Since you last donated plasma: Yes No 3. Female Donors: Have you been pregnant or are you pregnant now? 4. Have you had any new medical problems or diagnoses? 5. Have you had any new medical treatments, vaccinations or medications? 6. Have you had contact with someone who had a smallpox vaccination? 7. Have you donated whole blood, platelets or plasma at another center? Risk Activities Please review our Risk Poster Yes No |
| Changes in Health Since you last donated plasma: Yes No 3. Female Donors: Have you been pregnant or are you pregnant now? 4. Have you had any new medical problems or diagnoses? 5. Have you had any new medical treatments, vaccinations or medications? 6. Have you had contact with someone who had a smallpox vaccination? 7. Have you donated whole blood, platelets or plasma at another center? Risk Activities Please review our Risk Poster Yes No |
| Since you last donated plasma: Yes No 3. Female Donors: Have you been pregnant or are you pregnant now? 4. Have you had any new medical problems or diagnoses? 5. Have you had any new medical treatments, vaccinations or medications? 6. Have you had contact with someone who had a smallpox vaccination? 7. Have you donated whole blood, platelets or plasma at another center? Risk Activities Please review our Risk Poster Yes No |
| 3. Female Donors: Have you been pregnant or are you pregnant now? 4. Have you had any new medical problems or diagnoses? 5. Have you had any new medical treatments, vaccinations or medications? 6. Have you had contact with someone who had a smallpox vaccination? 7. Have you donated whole blood, platelets or plasma at another center? Risk Activities Please review our Risk Poster Yes No |
| you pregnant now? 4. Have you had any new medical problems or diagnoses? 5. Have you had any new medical treatments, vaccinations or medications? 6. Have you had contact with someone who had a smallpox vaccination? 7. Have you donated whole blood, platelets or plasma at another center? Risk Activities Please review our Risk Poster Yes No |
| 5. Have you had any new medical treatments, vaccinations or medications? 6. Have you had contact with someone who had a smallpox vaccination? 7. Have you donated whole blood, platelets or plasma at another center? Risk Activities Please review our Risk Poster Yes No |
| vaccinations or medications? 6. Have you had contact with someone who had a smallpox vaccination? 7. Have you donated whole blood, platelets or plasma at another center? Risk Activities Please review our Risk Poster Yes No |
| 7. Have you donated whole blood, platelets or plasma at another center? Risk Activities Please review our Risk Poster Yes No |
| another center? Risk Activities Please review our Risk Poster Yes No |
| Please review our Risk Poster Yes No |
| 8. Did you review the Risk Poster? |
| 9. Do you have any questions about anything mentioned on the Risk Poster? |
| 10. Since you last donated plasma, does anything on the Risk Poster apply to you? |
| Since you last donated plasma: Yes No |
| 11. Have you gotten a tattoo or had one touched up? |
| 12. Have you had an ear or body piercing? |

# PPTA Abbreviated Donor History Questionnaire For Frequent Plasma Donors

| | Yes No |
|---|---|
| <b>Optional Question A.</b> Have you had surgery oprocedure? | or a diagnostic, medical or dental |
| Optional Question B. Have you had acupunct | ture? |
| Additional Questions: | |
| Acknowledgment: | |
| I have reviewed the educational materials required transmitted by my donation, such as, Syphilis | s, HIV, Hepatitis B and C. |
| <ol><li>I agree not to donate if my donation could res<br/>receive plasma products.</li></ol> | sult in a potential risk to people who |
| 3. A sample of my blood will be tested for infect donation, such as, Syphilis, HIV, Hepatitis B | , , |
| <ol> <li>I understand you will attempt to notify me if for<br/>records will be maintained indicating the reas<br/>time period.</li> </ol> | • |
| <ol> <li>I have reviewed the information regarding the<br/>donating Source Plasma.</li> </ol> | e potential risks and hazards of |
| <ol> <li>I have been given the opportunity to ask question withdraw from the donation procedure at any</li> </ol> | <del>-</del> |
| Donor Signature: | Date: |

rBV A/B
Clinical Protocol IND 015155

# **APPENDIX E**

ADVERSE EVENT RECORDING SHEET FOR IDENTIFICATION OF POSSIBLE SERIOUS ADVERSE EVENTS (SAES)

# Tolerability and Immunogenicity of a Single 40-µg Dose of Recombinant Botulinum Vaccine A/B (rBV A/B) for the Production of BabyBIG® in Volunteers with Existing Botulinum Immunity

# Adverse Events Recording Sheet for Identification of Possible Serious Adverse Events (SAEs)

| Study Site/Location*:/ | | _ Participant S | Participant Study ID Number*: | |
|---|---|---|---|---|
| Participant Name: | | | | |
| Recombinant vaccine given: | Date: | | Time: | AM / PM |

- You may or may not experience any adverse events. The purpose of this recording sheet is for you to
  document at home any adverse events during the course of the study, if such should occur.
- If you make an error while recording, please draw a single line through the error, add your correction and initial. Please no white out or multiple lines through errors.
- The information you document on this form will be queried for by study staff during on-site study visits and phone call follow-up for safety at Weeks 1, 4, 10 and 26.
- Please indicate the date and time (if relevant) of each event's occurrence, as well as the date/time of the
  event's resolution.
- Please categorize the event's severity as indicated below.

**Note:** If you experience severe, life-threatening or any of the following neuromuscular symptoms (blurred or double vision, drooping of eyelids, drooping of the mouth, dry mouth, difficulty swallowing, difficulty speaking, weakness of an arm or leg, lack of coordination, shallow breathing, sensitivity to sunlight, or inability to perspire), **please seek** medical attention <u>immediately</u> and notify Dr. Khouri (24/7/365 phone # 925-408-5935) or Dr. Bloomfield (24/7/365 phone #: 614-595-5505) as soon as possible.

mild = you are able to perform all routine daily activities

moderate = you are able to perform some routine activities, but are limited in others severe = you are unable to perform all routine activities, often seeking medical care

| # | Reaction or Event<br>Description/Location | New<br>Event?<br>(Y/N) | Date /<br>Time<br>Started | Date /<br>Time<br>Ended | Severity | Treatment | Comments |
|---|---|---|---|---|---|---|---|
| | | / | / | | | | |
| | | / | | | | | |
| | / | | | | | | |

Additional Comments, if any (please continue on reverse side).

\* To be filled in by study staff

Ver. August 2018

Site Investigator's Initials\_\_\_\_\_

<sup>\*</sup>Please categorize the severity of the reaction as:

# Tolerability and Immunogenicity of a Single 40-µg Dose of Recombinant Botulinum Vaccine A/B (rBV A/B) for the Production of BabyBIG® in Volunteers with Existing Botulinum Immunity

# Adverse Events Recording Sheet for Identification of Possible Serious Adverse Events (SAEs)

| Study Site/Location*:// | Participant Study ID Number*: |
|-----------------------------------------|-----------------------------------|
| Additional Comments, if any: | |
| / | |
| Reviewed by: Site Principal Investigato | Date:// Time:AM/PM or or Designee |
| one i imopai investigate | r or Boolghoo |
| Title: | <u> </u> |
| * To be filled in by study staff | |
| Ver. August 2018 | Site Investigator's Initials |